# J2T-DM-KGAF Protocol (2)

A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Evaluate the Efficacy and Safety of Lebrikizumab in Patients With Moderate-to-Severe Atopic Dermatitis

NCT03443024

Approval Date: 07-MAR-2018



A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING TRIAL TO EVALUATE THE EFFICACY AND SAFETY OF LEBRIKIZUMAB IN PATIENTS WITH MODERATE-TO-SEVERE ATOPIC DERMATITIS

Protocol Number DRM06-AD01

Protocol Final Date 27 November 2017

Study Drug Lebrikizumab (DRM06)

**IND Number** 119866

Sponsor Dermira, Inc.

275 Middlefield Road Menlo Park, CA 94025

**USA** 

Amendment (1) Date 29 January 2018

Amendment (2) Date 07 March 2018

## **CONFIDENTIAL INFORMATION**

The information contained herein is confidential and the proprietary property of Dermira. Any use or disclosure of such information without the prior written authorization of Dermira is expressly prohibited.

# PROTOCOL AMENDMENT 2.0 (SUMMARY OF CHANGES)

The changes in the table below are new changes being introduced to Amendment 2.0. Additions are noted in **bold** and strikethroughs are as made. Minor corrections/additions may not be included.

| Section | Modified Text or Description | Rationale |
|---|---|---|
| 6.5 Study-Drug<br>Accountability | The Investigator must keep an accurate record of the number of cartons received, the study drug dispensed/used, and those returned to the Sponsor or designee. The Sponsor will provide forms to facilitate inventory control. All study-drug accountability forms and treatment logs must be retained in the Investigator's permanent study file, and these records must be available for inspection at any time by the Sponsor, its designees, or by regulatory agencies. | To accommodate sites with SOPs in place for destruction of unused study drug. |
| | The study monitor will perform drug accountability for all study drug at the site, and will assist in returning all used, unused, and expired study drug, to the Sponsor/designee, or verify study-drug destruction according to the study site's standard operating procedure, if it is accepted by the Sponsor.designee. | |
| 6.7 Study-Drug<br>Administration | Study drug is to be administered to all patients in the clinic by designated and trained study personnel. Study drug should be prepared in advance and injected subcutaneously according to the following instructions: | Feedback from investigators indicated that patients may |
| | <ul> <li>Remove study drug from refrigerated condition and<br/>allow to warm to room temperature for 15 minutes<br/>prior to administration. Study drug should be<br/>administered within 4 hours.</li> </ul> | prefer not having<br>4 injections given<br>at the same site. |
| | <ul> <li>Identify location for injections. Study drug may be injected in the abdomen, upper arm, or thigh. All injections administered at a single visit should be given in the same area, but may be split up into different areas for Week 0 and Week 2, which have 4 injections/visit. Injection sites should be ≥10 cm from one another. If possible, injections should not be administered at sites with active AD or other skin lesions.</li> </ul> | |
| | Inject study drug subcutaneously. | |
| | Record location of study injections in the eCRF. | |
| | <ul> <li>Properly dispose of used syringe according to site<br/>requirements. Syringe box must be kept for full drug<br/>accountability.</li> </ul> | |

| Section | Modified Text or Description | Rationale |
|---|---|---|
| 9.4. Laboratory<br>Evaluations | The inclusion of TB testing in Table 2 was not correct. It has been deleted from the table to make it consistent with the Schedule of Visits and Procedures in Appendix 1. | TB testing was not intended to be performed for this study. This oversight is being corrected with this amendment. |
| Appendix 1 | Add a checkbox for ECG assessment at Early termination visit | It was inadvertently left out. |
| Appendix 1 | Added collection of and procedure/therapy information. | It was inadvertently left out. |

# PROTOCOL AMENDMENT 1.0 (SUMMARY OF CHANGES)

The changes in the table below are new changes being introduced to Amendment 1.0. Additions are noted in **bold** and strikethroughs are as made. Minor corrections/additions may not be included.

| Section | Modified Text or Description | Rationale |
|---|---|---|
| 6.4. Study-Drug<br>Unblinding | The Sponsor or designee, the Investigator, study-site personnel, and the patient will be blinded to treatment assignment. The integrity of the clinical study will be maintained by observing the treatment blind. If knowledge of a patient's treatment assignment is required for the patient's clinical care and/or safety, the Investigator will open the Code-Breaking Card received with the study-drug kit. The Code-Breaking Card should be stored in a secure, locked location at the site. The Investigator should have access to the Code-Breaking Card at all times (e.g., 24/7). is permitted to use the IWRS to obtain treatment assignment. The Investigator should consult with the Sponsor's medical monitor prior to obtaining treatment assignment information. The Investigator must document (in the patient's medical record) the date and time the blind was broken, the names of the personnel involved, and the reason that treatment assignment information was required. | Because of the secondary packaging used for the kits in this study, the CRO was unable to accommodate use of an IWRS system. Instead, in the event of an unblinding, Code-Breaking Cards will be used. |
| 6.7. Study-Drug<br>Administration | Study drug is to be administered to all patients in the clinic by designated and trained study personnel. Study drug should be prepared in advance and injected subcutaneously according to the following instructions: Remove study drug from refrigerated condition and allow to warm to room temperature for 15 minutes prior to administration. Study drug should be administered within 4 hours. | Change of procedure. Sites will dispose of syringes instead of returning them to the carton. Study drug should not be left at room |
| | <ul> <li>Identify location for injections. Study drug may be injected in the abdomen, upper arm, or thigh. All injections administered at a single visit should be given in the same area. Injection sites should be ≥10 cm from one another. If possible, injections should not be administered at sites with active AD or other skin lesions.</li> </ul> | temperature for longer than 4 hours. |
| | Inject study drug subcutaneously. | |
| | Record location of study injections in the eCRF. | |
| | <ul> <li>Properly dispose of used syringe according to<br/>site requirements. Syringe box must be kept for<br/>full drug accountability.</li> </ul> | |

| Section | Mc | odified Text or Description | Rationale |
|---|---|---|---|
| 7.2. Baseline Visit | • | Confirm emollient use. | Tablet will be |
| (Day 1) | • | Re-assess and confirm patient eligibility (Inclusion/Exclusion criteria). | dispensed at Baseline visit, not at Screening visit. |
| | • | Measure weight and vital signs. | at Screening visit. |
| | • | Collect concomitant medication information. | |
| | • | Query for adverse events (AEs) since the last visit. | |
| | • | Collect a 12-lead ECG. | |
| | • | Draw blood samples for laboratory tests (hematology and chemistry) | |
| | • | Draw a pre-dose blood sample for PK and anti-drug antibody (ADA) testing. | |
| | • | Conduct urine for urinalysis and urine pregnancy test (WOCBP only). | |
| | • | Dispense electronic tablet that will be used for daily home recording of pruritus NRS, sleep-loss NRS, and ADIQ. | |
| | • | Train patient on the use of the electronic tablet. | |
| | • | Review compliance report on the electronic tablet for the daily assessments (pruritus NRS, sleep-loss NRS, and ADIQ) and remind patient to continue daily record. | |
| | • | Complete the following assessments: | |
| | | <ul> <li>Investigator's Global Assessment (IGA)</li> </ul> | |
| | | <ul> <li>Eczema Area and Severity Index (EASI)</li> </ul> | |
| | | <ul> <li>Body Surface Area (BSA)</li> </ul> | |
| | | <ul> <li>Patient Oriented Eczema Measure (POEM)</li> </ul> | |
| | | <ul> <li>Dermatology Life Quality Index (DLQI)</li> </ul> | |
| | | <ul> <li>Hospital Anxiety and Depression Scale (HADS)</li> </ul> | |
| | • | Randomize the patient. | |
| | • | Administer study drug. | |
| | • | Instruct the patient to apply an emollient twice daily. | |
| | • | Schedule next visit. | |

| Section | Modified Text or Description | Rationale |
|---|---|---|
| 11.6. Exposure and Compliance | The extent of exposure to study drug in each treatment group will be summarized by total number of days of exposure, total number of applications, number of missed applications, and number and percentage of patients who are compliant. An application is considered the full set of injections (either 2 or 4 depending on visit) specified by the protocol. | Clarification |
| | A patient will be considered compliant with the dosing regimen if the patient received ≥75% of the expected number of applications while enrolled in the study. | |
| Appendix 1. | Changed D224 to <b>D225</b> | Changes to |
| Schedule of Visits and Procedures | Noted that urine pregnancy test is for WOCBP only | reconcile the<br>Schedule of Visits<br>and Procedures |
| | Added DLQI, HADS, and Global Assessment of<br>Change to Early-Termination visit. | with the Study<br>Procedures |
| Appendix 5. Body<br>Surface Area<br>(BSA) | The BSA assessment estimates the extent of disease or skin involvement with respect to AD and is expressed as a percentage of total body surface. | BSA scores adjusted to sum to 100%. |
| | Determine BSA using the patient's palm = 1% rule. | |
| | The patient's palm is measured from the wrist to the proximal interphalangeal (PIP) and thumb. | |
| | Estimate the number of palms it takes to cover the affected AD area. Add up the number of palms to give a total estimate of the area covered in AD. | |
| | Below are estimates when entire areas (anterior and posterior) are covered: | |
| | Head and Neck = 10% (10 palms) | |
| | Upper Extremities = 20% (20 palms) | |
| | Trunk (axillae and groin) = 4030% (4030 palms) | |
| | Lower extremities (buttocks) = 40% (40 palms) | |

# A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING TRIAL TO EVALUATE THE EFFICACY AND SAFETY OF LEBRIKIZUMAB IN PATIENTS WITH MODERATE-TO-SEVERE ATOPIC DERMATITIS

## **CRO Personnel**



# **SAE/ Emergency Contact Information**



## **Sponsor Personnel**



## SPONSOR SIGNATURE PAGE

A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING TRIAL TO EVALUATE THE EFFICACY AND SAFETY OF LEBRIKIZUMAB IN PATIENTS WITH MODERATE-TO-SEVERE ATOPIC DERMATITIS

Protocol Number DRM06-AD01

Protocol Final Date 27 November 2017

Amendment (1) Date 29 January 2018

Amendment (2) Date 07 March 2018

The signature below constitutes approval of this protocol. I certify that I have the authority to approve this protocol on behalf of the Sponsor, Dermira, Inc. The study will be conducted in accordance with this protocol and all applicable laws, rules, and regulations and International Conference on Harmonization Good Clinical Practice (ICH GCP), regulations of the United States (US) Food and Drug Administration (FDA), and the ethical principles that have their origin in the Declaration of Helsinki.

| Authorized by: | |
|---------------------------------------------|-------------|
| PPD | |
| | 07 MAR ZOIF |
| Sponsor Signature | Date |
| PPD | |
| Senior Vice President, Clinical Development | |

DRM06-AD01-A2

## **INVESTIGATOR SIGNATURE PAGE**

I have read this protocol, including the appendices, and agree that it contains all necessary details for carrying out the study as described. I will conduct this protocol as outlined herein, according to the ethical principles that have their origin in the Declaration of Helsinki, International Conference on Harmonization (ICH) guidelines for Good Clinical Practice (GCP) and applicable laws, rules and regulatory requirement(s) including those of the United States (US) Food and Drug Administration (FDA).

I agree to obtain the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval of the protocol and informed consent prior to the start of the study.

I agree to obtain formal written informed consent in accordance with applicable federal and local regulations and international guidelines from all patients prior to their entry into the study.

I have received and reviewed the Investigator's Brochure including the potential risks and side effects of the product and instructions for use.

I agree to report to the Sponsor any adverse events that occur during the study in accordance with the ICH GCP guideline and the protocol.

I agree to ensure that all associates, colleagues, and employees assisting me with the conduct of the study are informed of their responsibilities in meeting the above commitments and the commitments set forth in the Investigator's Agreement.

I agree to maintain adequate and accurate records and to make those records available for inspection in accordance with the ICH GCP guideline, and federal and local requirements.

I understand that the study may be terminated or enrollment suspended at any time by the Sponsor, with or without cause, or by me if it becomes necessary to protect the best interests of the study patients.

| Investigator's Signature | Date |
|-----------------------------|------|
| Investigator's Name (print) | |

## **PROTOCOL SYNOPSIS**

| Title: | A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Evaluate the Efficacy and Safety of Lebrikizumab in Patients with Moderate-to-Severe Atopic Dermatitis |
|---|---|
| Protocol Number: | DRM06-AD01 |
| Phase: | 2b |
| Number of Sites: | Approximately 60 in the United States |

## **Study Population:**

Patients with moderate-to-severe atopic dermatitis (AD) who are candidates for systemic therapy.

## Sample Size:

Approximately 275

## **Study Objectives:**

- To evaluate the safety and efficacy of lebrikizumab compared with placebo in patients with moderate-to-severe AD.
- To evaluate the dose-response of lebrikizumab in patients with moderate-to-severe AD.

## **Duration of Patient Participation:**

- Screening: Maximum duration of 30 days;
- Treatment period: Approximately 113 days
- Post-treatment follow-up period: Approximately 111 days
- Maximum total participation: Approximately 257 days

#### **Study Treatment:**

Lebrikizumab, 125 mg/mL injectable delivered in a pre-filled syringe (PFS) Placebo. 0 mg/mL injectable delivered in a PFS

## Study Design:

This is a randomized, double-blind, placebo-controlled, parallel-group study. Approximately 275 patients with moderate-to-severe AD will be enrolled into this 32-week study.

Patients will be seen every two weeks and receive all study drug injections in the clinic. Patients will be evaluated for safety and efficacy through Week 16 on study. A safety follow-up visit will occur at Week 24 and a follow-up phone call will occur at Week 32.

Serum PK and anti-drug antibody (ADA) will be collected from all patients. PK samples will be collected at Baseline, Weeks 2, 4, 8, 12, 16, and 24. ADA samples will be collected at Baseline, Weeks 2, 4, 16, and 24.

Patients will be randomized 3:3:3:2 to the following treatment groups.

## Treatment Group 1: Lebrikizumab, 125 mg every 4 weeks

Baseline: Loading dose of 250 mg (2 injections of 1 mL of 125 mg/mL drug product and 2 injections of 1-mL placebo)

Week 2: Four 1-mL injections of placebo

Weeks 4, 8, 12: 125 mg (one 1-mL injection of 125 mg/mL drug product and one 1-mL injection of placebo)

Weeks 6, 10, 14: Two 1-mL injections of placebo

Treatment Group 2: Lebrikizumab, 250 mg every 4 weeks

Baseline: Loading dose of 500 mg (four 1-mL injections of 125 mg/mL drug product)

Week 2: Four 1-mL injections of placebo

Weeks 4, 8, 12: 250 mg (two 1-mL injections of 125 mg/mL drug product)

Weeks 6, 10, 14: Two 1-mL injections of placebo

Treatment Group 3: Lebrikizumab, 250 mg every 2 weeks

Baseline and Week 2: Loading dose of 500 mg (four 1-mL injections of 125 mg/mL drug product)

Week 4, 6, 8, 10, 12, 14: 250 mg (two 1-mL injections of 125 mg/mL drug product)

Treatment Group 4: Placebo every 2 weeks

Baseline and Week 2: Four 1-mL injections of placebo

Week 4, 6, 8, 10, 12, 14: Two 1-mL injections of placebo

## **Key Inclusion Criteria:**

- Male or female, 18 years or older.
- Chronic AD as defined by Hanifin and Rajka (1980) that has been present for ≥1 year before the screening visit (see Appendix 2)
- Eczema Area and Severity Index (EASI) score ≥16 at the screening and the Baseline visit.
- Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the screening and the Baseline visit.
- ≥10% body surface area (BSA) of AD involvement at the screening and the Baseline visit.

#### **Kev Exclusion Criteria:**

- Treatment with any of the following agents within 4 weeks prior to the Baseline visit:
  - Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
  - Phototherapy and photochemotherapy (PUVA) for AD.
- Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 1 week prior to the Baseline visit.
- Treatment with:
  - An investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, prior to the Baseline visit.
  - Dupilumab within 3 months prior to Baseline visit.
  - Cell-depleting biologics, including rituximab, within 6 months prior to the Baseline visit.
  - Other biologics within 5 half-lives (if known) or 16 weeks prior to Baseline visit (whichever is longer).

• Use of prescription moisturizers within 7 days of the Baseline visit.

## **Primary Endpoint:**

• Percent change in Eczema Area and Severity Index (EASI) from Baseline to Week 16.

## **Secondary Endpoints:**

- Proportion of patients with a 75% improvement from Baseline in EASI (EASI75) at Week 16.
- Proportion of patient with an IGA score of 0 (clear) or 1 (almost clear) and a reduction ≥2 points from Baseline to Week 16 (5-point scale).
- Proportion of patients with EASI <7 at Week 16.
- Proportion of patients achieving EASI50 and EASI90 at Week 16.
- Percent change in the sleep-loss numerical rating scale (NRS) score from Baseline to Week 16.
- Percent change in pruritus NRS score from Baseline to Week 16.
- Proportion of patients with pruritus NRS change of ≥3 from Baseline to Week 16.
- Proportion of patients with pruritus NRS change of ≥4 from Baseline to Week 16.
- Change in Body Surface Area (BSA) involved with AD from Baseline to Week 16.
- Change from Baseline in Atopic Dermatitis Impact Questionnaire (ADIQ) score.

# **TABLE OF CONTENTS**

| <b>PROTO</b> | COL AMENDMENT 2.0 (SUMMARY OF CHANGES) | 2 |
|---|---|---|
| | COL AMENDMENT 1.0 (SUMMARY OF CHANGES) | |
| | OR SIGNATURE PAGE | |
| INVESTI | GATOR SIGNATURE PAGE | ç |
| | COL SYNOPSIS | |
| | OF CONTENTS | |
| | TABLES | |
| | APPENDICES | |
| | BACKGROUND | |
| <b>1</b><br>1.1 | Atopic Dermatitis | |
| 1.1 | Lebrikizumab | |
| 1.3 | Study Rationale and Benefit-Risk Assessment | |
| 1.3.1 | Scientific Rationale: Evidence of the Role of IL-13 in AD | |
| 1.3.2 | Summary of Clinical Development | |
| 1.3.2.1 | Efficacy | |
| 1.3.2.2 | Safety | |
| 1.4<br>1.5 | Rationale for Treatment Regimen | |
| 2 | STUDY OBJECTIVES | |
| 3 | STUDY ENDPOINTS | |
| 3.1<br>3.2 | Primary Endpoint: Secondary Endpoints: | |
| 3.2<br><b>4</b> | STUDY DESIGN | |
| <b>4</b><br>4.1 | Duration of the Study | |
| 4.2 | Study Population and Number of Patients | |
| 5 | SELECTION OF PATIENTS | |
| 5.1 | Inclusion Criteria | |
| 5.2 | Exclusion Criteria | |
| 6 | STUDY DRUG. | 23 |
| 6.1 | Study-Drug Formulation and Presentation | 23 |
| 6.2 | Study-Drug Supply and Labeling | |
| 6.3 | Study-Drug Storage | |
| 6.4 | Study Drug Assouptshility | |
| 6.5<br>6.6 | Study-Drug Accountability Patient Randomization | |
| 6.7 | Study-Drug Administration | |
| 6.8 | Concomitant Medications and Procedures | |
| 6.9 | Permitted and Prohibited Treatments and Procedures | 26 |
| 6.10 | Rescue Therapy | 26 |
| 7 | Study PROCEDURES | |
| 7.1 | Screening Visit | |
| 7.2 | Baseline Visit (Day 1) | |
| 7.3<br>7.4 | Visits on Day 15, Day 29, Day 43, Day 57, Day 71, Day 85 and Day 99 (+/- 3 Day) | |
| 7.4<br>7.5 | Visit Day 113 (Week 16) (+/- 3 Day) (End-of-Treatment/Early-Termination Visit) Follow-Up Visit Day 141 (Week 20) (+/- 7 Days) | |
| 7.6 | Follow-Up Visit Day 141 (Week 24) (+/- 7 Days) | |

| 7.7 | Follow-Up Visit Phone Call, Day 225 (Week 32) (+/- 7 Days) | 30 |
|---|---|---|
| 7.8 | Unscheduled Visits | 30 |
| 8 | DETAILS OF ASSESSMENTS | 30 |
| 8.1 | Screening Assessments | 30 |
| 8.1.1 | Demographics | |
| 8.1.2 | Medical History | |
| 8.1.3 | Disease Specific Information | |
| 8.2 | Assessment of Efficacy | |
| 8.2.1 | AD Assessments | |
| 8.2.1.1 | Investigator Global Assessment (IGA) | |
| 8.2.1.2 | Eczema Area and Severity Index (EASI) | |
| 8.2.1.3 | Body Surface Area (BSA) | |
| 8.2.1.4 | Pruritus | |
| 8.2.1.5 | Sleep-Loss | |
| 8.2.1.6 | Atopic Dermatitis Impact Questionnaire (ADIQ) | |
| 8.2.1.7 | Patient Oriented Eczema Measure (POEM) | |
| 8.2.1.8 | Dermatology Life Quality Index (DLQI) | |
| 8.2.1.9 | Hospital Anxiety and Depression Scale (HADS) | |
| | Global Assessment of Change–AD | |
| 8.2.2 | PK and ADA Sampling | |
| 9 | ASSESSMENT OF SAFETY | |
| 9.1 | Assessment of Safety | |
| 9.1.1 | Physical Examination | |
| 9.1.2 | Vital Signs | |
| 9.1.3 | ECGs | |
| 9.1.4 | Laboratory Evaluations | |
| 9.1.5 | Adverse Events (AEs) | |
| 9.1.5.1<br>9.1.6 | Reporting | |
| 9.1.6<br>9.1.6.1 | Serious Adverse Events (SAEs) | |
| 9.1.0.1 | Adverse Events of Special Interest (AESI) | |
| 9.1.8 | Pregnancy | |
| <b>10</b> | STUDY DISCONTINUATIONS | |
| 10.1 | Study Termination Early Termination of Study Patients | |
| 10.2<br>10.3 | Study-Drug Discontinuation | |
| 11 | STATISTICAL CONSIDERATIONS | |
| 11.1 | General Statistical Methodology | |
| 11.2 | Populations Analyzed | |
| 11.3<br>11.4 | Primary Efficacy | |
| 11. <del>4</del><br>11.5 | Secondary Efficacy | |
| 11.6 | PK Analysis Exposure and Compliance | |
| 11.6 | Adverse Events | |
| 11.7 | Other Safety Data | |
| 11.0 | Sample-Size Determination. | |
| | • | |
| <b>12</b> | ADMINISTRATION | |
| 12.1<br>12.2 | Compliance with the Protocol | |
| 12.2 | Informed Consent Procedures | |
| 14.J | OLUMY DOCUMENTATION AND THE CONF | 44 |

| Lebrikizumab DRM06 | | DRM06-AD01-A2 |
|---|---|---|
| 12.4 St | udy Monitoring | 42 |
| | tention of Study Documentation | |
| 12.6 Ac | ronyms | 43 |
| 13 RI | FERENCES | 45 |
| 14 AI | PPENDICES | 48 |
| LIST OF TA | ABLES | |
| Table 1 | Dosing Schedule by Treatment Group | 25 |
| Table 2 | Laboratory Parameters | 34 |
| LIST OF AI | PPENDICES | |
| Appendix 1 | Schedule of Visits and Procedures | 48 |
| Appendix 2 | Hanifin/Rajka Diagnostic Criteria for Atopic Dermatitis | 50 |
| Appendix 3 | Investigator Global Assessment (IGA) | 51 |
| Appendix 4 | Eczema Area and Severity Index (EASI) | 52 |
| Appendix 5 | | |
| Appendix 6 | Pruritus Numeric Rating Scale (NRS) | 54 |
| Appendix 7 | | |
| Appendix 8 | • | |
| Appendix 9 | | |
| Appendix 1 | | |
| Appendix 1 | | |
| Appendix 1 | | |

#### 1 BACKGROUND

#### 1.1 Atopic Dermatitis

Atopic dermatitis (AD) is a relapsing and remitting inflammatory skin disorder that affects all age groups. It is chronic and incurable, and is characterized by skin-barrier disruption and immune dysregulation (largely mediated by type-2 helper T cells). Clinically, AD is characterized by xerosis, erythematous crusted eruption (dermatosis), lichenification, an impaired skin barrier, and intense pruritus. AD flares are frequently triggered by exposure to environmental factors, irritants, and allergens.

Although estimates of AD prevalence vary widely across different studies due to differences in data collection methodology, inconsistent age group assessment, and study periods, AD is one of the most common dermatologic diseases—15–30% of children and 2–10% of adults are affected, and prevalence appears to have increased over the past two to three decades. There appears to be some geographic variability in prevalence. Prevalence in children has been estimated to be 5.9–16.0% in Western Europe and 10.7% in the United States (US)<sup>5,6</sup> In adults, prevalence has been reported as 0.3–2.0% in Europe, 4.9% in the United Kingdom (UK), and 2.4–6.0% in the US. With respect to disease severity, 14% of AD patients in the UK have moderate disease and 2% have severe disease. A recent US study measuring AD severity in children found that for 67% disease was mild, for 26% it was moderate, and for 7% it was severe. Approximately 85% of all cases of AD begin before age 5, with up to 70% of children having spontaneous remission before adolescence.

Patients with AD have a high disease burden and their quality of life (QoL) is significantly affected. In one study, AD was shown to have a greater negative effect on patient mental health than diabetes and hypertension. <sup>10</sup> Patients with moderate-to-severe AD have a higher prevalence of social dysfunction and sleep impairment, which are directly related to the severity of the disease. <sup>4</sup> Depression, anxiety, and social dysfunction not only affect patients with AD, but also affect their caregivers. <sup>10</sup> Compared with psoriasis, another common and debilitating skin disease, patients with AD have lower physical vitality, social functioning, role-emotional, and mental health scores. <sup>11</sup>

The therapeutic approach to AD primarily consists of trigger avoidance, skin hydration with bathing, and use of emollients and anti-inflammatory therapies consisting predominantly of topical corticosteroids (TCS). In many patients, treatment with TCS provides some measure of symptomatic relief but does not adequately control the disease.

In those patients who have persistent moderate-to-severe disease not responding adequately to TCS, guidelines outline several step-up therapeutic options. The step-up options include topical calcineurin inhibitors (TCIs), phototherapy, and immunosuppressive agents such as oral corticosteroids, cyclosporine, azathioprine, methotrexate, and mycophenolate mofetil. Among these, only cyclosporine is approved for treatment of moderate-to-severe AD (nationally licensed in many European countries, but not in the U.S.), and its use is limited to patients  $\geq$ 16 years for a maximum treatment period of 8 weeks (Neoral®). Recently, the anti-IL-4R agent, dupilimab, was approved for the treatment of moderate-to-severe AD. Dupilimab's mechanism of action is likely through inhibition of heterodimerization of the IL-4R $\alpha$ /IL-13R $\alpha$ 1 complex, preventing IL-13 from initiating downstream signaling through the JAK/STAT pathway.

## 1.2 Lebrikizumab

Lebrikizumab is a humanized monoclonal immunoglobulin (Ig) G4 antibody (hulgG4) with a mutation in the hinge region for increased stability. Lebrikizumab binds specifically to soluble human interleukin (IL)-13 with high affinity, and potently inhibits IL-13 signaling through the IL-4R $\alpha$ /IL-13R $\alpha$ 1 complex. Because lebrikizumab binds to IL-13 in a non-receptor binding domain (i.e., a portion of the molecule not involved in binding to its receptor), antibody-bound IL-13 can still bind its receptor (IL-13 R $\alpha$ 1), but the receptor complex is not activated.

Because lebrikizumab does not bind to IL-13 in mice, the most commonly used species for animal models of AD, it was not possible to perform in vivo lebrikizumab pharmacology or efficacy studies in an animal model of AD. However, several non-clinical studies in the literature demonstrate increased expression of IL-13 in affected skin, supporting the use of an anti-IL-13 therapeutic for human AD.

Two previous studies were conducted with lebrikizumab in patients with AD. They are described in Section 1.3.2. See the Lebrikizumab Investigator's Brochure (IB) for additional details on lebrikizumab non-clinical and clinical studies.

## 1.3 Study Rationale and Benefit-Risk Assessment

## 1.3.1 Scientific Rationale: Evidence of the Role of IL-13 in AD

AD is a T-helper type 2 (Th-2)-driven inflammatory disease. Several lines of evidence from published literature implicate IL-13 as a key component of AD pathobiology:

- Genetic studies have shown that polymorphisms in the gene for IL-13,<sup>14, 15</sup> and in the IL-4Rα receptor<sup>16</sup> are associated with an increased risk for developing AD.
- IL-13 can act on keratinocytes in the skin to downregulate their differentiation; <sup>17</sup> and to induce T-cell chemoattractants that mediate T cell infiltration into AD lesions. <sup>18</sup>
- II-13 may induce IL-5 expression and eosinophil infiltration through the induction of eosinophil chemoattractants.<sup>19</sup>
- IL-13 can reduce epithelial integrity through the downregulation of filaggrin, loricrin, and involucrin.<sup>20</sup>
- IL-13 can mediate fibrosis through the induction of collagen production in fibroblasts.<sup>21</sup>
- In an epi-cutaneous ovalbumin sensitization model of murine AD, topical anti-sense oligonucleotides targeting mouse IL-13 mRNA were shown to significantly reduce the production of IL-13 in the skin and in turn significantly reduce inflammation.<sup>22</sup>
- Increased IL-13 has been reported in the serum of AD patients<sup>16</sup> and several studies have reported an increase in IL-13 expressing T cells in the blood of AD patients.<sup>23-25</sup>
- Increased expression of IL-13 in AD skin has been reported.<sup>26-31</sup>
- Increased levels of IL-13 have been observed in AD skin lesions and reports suggest a relationship between IL-13 expression and the severity of disease.<sup>25</sup>
- Clinical studies investigating agents with broadly acting anti-inflammatory activity demonstrated that reduced IL-13 expression was associated with clinical improvement.<sup>32-34</sup>

- Clinical studies with two monoclonal antibodies (tralokinumab and dupilimab) that inhibit IL-13 demonstrated clinical benefit to patients with AD. Tralokinumab, an anti-IL-13 monoclonal antibody, was tested in combination with TCS.<sup>35</sup> Dupilimab, an anti-IL4R agent that inhibits the activity of IL-13 by preventing heterodimerization of the 4Rα/IL-13Rα1 complex, was efficacious as a monotherapy or in combination with TCS.<sup>36</sup>
- Data from a Phase 2a study with lebrikizumab CCI demonstrated clinical benefit in patients with AD.

## 1.3.2 Summary of Clinical Development

Two clinical studies of lebrikizumab in AD have been performed.



## 1.3.2.1 Efficacy





# 1.3.2.2 Safety



# 1.4 Rationale for Treatment Regimen



# 1.5 Study Conduct Statement

This study will be conducted in compliance with the protocol, according to current United States federal regulations (21, Code of Federal Regulations [CFR] Parts 50, 56 and 312D) and the principles of International Conference on Harmonization (ICH) (ICH E6[R2]-June 2015) Good Clinical Practice (GCP), Food and Drug Administration (FDA) guidelines and the Declaration of Helsinki, 1964 (as amended in Edinburgh [2000]).

#### 2 STUDY OBJECTIVES

To evaluate the safety and efficacy of lebrikizumab compared with placebo in patients with moderate-to-severe AD.

To evaluate the dose-response of lebrikizumab in patients with moderate-to-severe AD.

## 3 STUDY ENDPOINTS

## 3.1 Primary Endpoint:

Percent change in Eczema Area and Severity Index (EASI) from Baseline to Week 16.

## 3.2 Secondary Endpoints:

- Proportion of patients with a 75% improvement from Baseline in EASI (EASI75) at Week 16.
- Proportion of patient with an IGA score of 0 (clear) or 1 (almost clear) and a reduction
   ≥2 points from Baseline to Week 16 (5-point scale, 0–4).
- Proportion of patients with EASI <7 at Week 16.
- Proportion of patients achieving EASI50 and EASI90 at Week 16.
- Percent change in the sleep-loss numerical rating scale (NRS) score from Baseline to Week 16.
- Percent change in pruritus NRS score from Baseline to Week 16.
- Proportion of patients with pruritus NRS change of ≥3 from Baseline to Week 16.
- Proportion of patients with pruritus NRS change of ≥4 from Baseline to Week 16.
- Change in Body Surface Area (BSA) involved with AD from Baseline to Week 16.
- Change from Baseline in ADIQ score.

## 4 STUDY DESIGN

#### 4.1 Duration of the Study

The screening period will be no more than 30 days. The treatment period will be from Baseline to Week 16 (113 days). The follow-up period will last through Week 32. The maximum total participation is approximately 257 days.

## 4.2 Study Population and Number of Patients

Approximately 275 patients, ≥18 years, will be enrolled.

## 5 SELECTION OF PATIENTS

#### 5.1 Inclusion Criteria

Patients must meet all the following criteria to be eligible for this study:

- 1. Male or female, ≥18 years.
- 2. Chronic AD as defined by Hanifin and Rajka (1980) that has been present for ≥1 year before the screening visit (see Appendix 2).
- 3. Eczema Area and Severity Index (EASI) score ≥16 at the screening and the Baseline visits.
- Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the screening and the Baseline visits.
- 5. ≥10% body surface area (BSA) of AD involvement at the screening and the Baseline visits.
- 6. History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable (e.g., because of important side effects or safety risks).
- 7. Applied a stable dose of topical emollient (over-the-counter moisturizer) twice daily for ≥7days prior to the Baseline visit.
- 8. Willing and able to comply with all clinic visits and study-related procedures and questionnaires.
- 9. Provide signed informed consent.

#### 5.2 Exclusion Criteria

Patients meeting any of the criteria below are not for this study:

- 1. History of anaphylaxis.
- 2. Participation in a prior lebrikizumab clinical study.
- 3. Treatment with any of the following agents within 4 weeks prior to the Baseline visit:
  - a. Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
  - b. Phototherapy and photochemotherapy (PUVA) for AD.
- 4. Treatment with TCS or TCI within 1 week prior to the Baseline visit.
- 5. Treatment with biologics as follows:
  - a. Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, prior to the Baseline visit.
  - b. Dupilimab within 3 months of Baseline visit.
  - c. Cell-depleting biologics, including to rituximab, within 6 months prior to the Baseline visit.
  - d. Biologics within 5 half-lives (if known) or 16 weeks prior to Baseline visit, whichever is longer.

- 6. Use of prescription moisturizers within 7 days of the Baseline visit.
- 7. Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the screening visit.
- 8. Treatment with a live (attenuated) vaccine within 12 weeks before the Baseline visit.
- 9. Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the Baseline visit, or superficial skin infections within 1 week before the Baseline visit. NOTE: patients may be rescreened after infection resolves.
- 10. Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., tuberculosis [TB], histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per the Investigator's judgment.
- 11. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
- 12. Positive with hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody at the screening visit.
- 13. In the Investigator's opinion, any clinically significant laboratory results from the chemistry, hematology or urinalysis tests obtained at the screening visit.
- 14. Presence of skin comorbidities that may interfere with study assessments.
- 15. History of malignancy within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
- 16. Severe concomitant illness(es) that in the Investigator's judgment would adversely affect the patient's participation in the study. Any other medical or psychological condition (including relevant laboratory abnormalities at screening) that in the opinion of the Investigator may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study patient because of his/her participation in this clinical trial, may make patient's participation unreliable, or may interfere with study assessments. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.
- 17. Women of reproductive potential\* who are sexually active and unwilling to use adequate birth control. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception<sup>†</sup> throughout the duration of the study and for 120 days after last dose of study drug.
- \*The following are considered women who are NOT of reproductive potential: Menopausal women, defined as ≥12 consecutive months without menses (if in question, a follicle stimulating hormone level of ≥25 mU/mL); Women surgically sterilized (history of hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).

<sup>†</sup>Includes abstinence, oral/implant/injectable/transdermal hormonal contraceptives, intrauterine device, double-barrier contraception (i.e., condom+diaphragm), same sex partner, or a male partner with vasectomy.

## 6 STUDY DRUG

## 6.1 Study-Drug Formulation and Presentation

The study drug used in this trial will be lebrikizumab and placebo. Lebrikizumab is a sterile liquid solution containing 125 mg/mL lebrikizumab, Placebo solution is identical in appearance and content to the active solution with the exception of lebrikizumab. All study drug will be supplied as a sterile pre-filled syringe with a pre-assembled needle safety device.

Each prefilled syringe is intended for a single-dose subcutaneous (SC) administration only.

## 6.2 Study-Drug Supply and Labeling

All study drug will be supplied as a sterile pre-filled syringe (PFS) with a pre-assembled needle safety device. Each PFS will be packaged in a syringe-box.

Pre-filled syringes will be labeled and will contain the pre-printed medication number (MEDNO), along with study drug storage instructions. The syringe-box label will also contain the corresponding pre-printed MEDNO and use by date, along with study-drug storage instructions. In addition, the syringe-box label will contain a write-in space for the patient number, investigator number and administration date. All labels will state "limited by U.S. law to investigational use".

Syringes and syringe boxes will be packaged in a secondary kit and labeled with a Kit Number. Kit Numbers will be assigned to a patient in the interactive web response system (IWRS) based on the study randomization schema.

## 6.3 Study-Drug Storage

Study drug is to be stored under refrigerated conditions (2–8°C) and protected from excessive light and heat. Study drug should not be frozen, shaken, or stored at room temperature.

Temperature excursions outside of 2–8°C must be reported to the Sponsor or the designee.

## 6.4 Study-Drug Unblinding

The Sponsor or designee, the Investigator, study-site personnel, and the patient will be blinded to treatment assignment. The integrity of the clinical study will be maintained by observing the treatment blind. If knowledge of a patient's treatment assignment is required for the patient's clinical care and/or safety, the Investigator will open the Code Breaking Card received with the study-drug kit. The Code-Breaking Card should be stored in a secure, locked location at the site. The Investigator should have access to the Code-Breaking Card at all times (e.g., 24/7). The Investigator should consult with the Sponsor's medical monitor prior to obtaining treatment assignment information. The Investigator must document (in the patient's medical record) the date and time the blind was broken, the names of the personnel involved, and the reason that treatment assignment information was required.

## 6.5 Study-Drug Accountability

The Investigator must keep an accurate record of the number of cartons received, the study drug dispensed/used, and those returned to the Sponsor or designee. The Sponsor will provide forms to facilitate inventory control. All study-drug accountability forms and treatment logs must be retained in the Investigator's permanent study file, and these records must be available for inspection at any time by the Sponsor, its designees, or by regulatory agencies.

The study monitor will perform drug accountability for all study drug at the site, and will assist in returning all used, unused, and expired study drug, to the Sponsor/designees, or destroy it according to the study site's standard operating procedure, if accepted by the Sponsor.

#### 6.6 Patient Randomization

All patients will be randomized to study treatment using an IWRS. Study randomization will occur across study sites. After written informed consent has been obtained, all patients will receive a six-digit screening number (XXX-XXX = site number-patient number), assigned in EDC (via iMedidata Rave in sequential order), which will be assigned by the site. Sites should assign the patient numbers in the order that they are screened and enter patients in EDC in the same order. Following completion of the screening period, and after all patient eligibility requirements are confirmed on Day 1 (Baseline), the patient's screening number will be entered in the IWRS, and the patient will be assigned a patient study-drug kit. One kit will provide all the study drug for that patient based on the assigned treatment group.

Patients will be randomized 3:3:3:2 to one of the following treatment groups. The dosing schedule by treatment group is shown in Table 1.

## Treatment Group 1: Lebrikizumab, 125 mg every 4 weeks

**Baseline:** Loading dose of 250 mg (two injections of 1 mL of 125 mg/mL drug product and two injections of 1 mL placebo);

Week 2: Four 1-mL injections of placebo

**Weeks 4, 8, 12:** 125 mg (one 1-mL injection of 125 mg/mL drug product and one 1-mL injection of placebo)

Week 6, 10, 14: Two 1-mL injections of placebo

## Treatment Group 2: Lebrikizumab, 250 mg every 4 weeks

**Baseline:** Loading dose of 500 mg (four 1-mL injections of 125 mg/mL drug product)

Week 2: Four 1-mL injections of placebo

Weeks 4, 8, 12: 250 mg (two 1-mL injections of 125 mg/mL drug product);

Week 6, 10, 14: Two 1-mL injections of placebo

### **Treatment Group 3**: Lebrikizumab, 250 mg every 2 weeks

**Baseline and Week 2:** Loading dose of 500 mg (four 1-mL injections of 125 mg/mL drug product)

Week 4, 6, 8, 10, 12, 14: 250 mg (two 1-mL injections of 125 mg/mL drug product)

## **Treatment Group 4:** Placebo every 2 weeks

**Baseline and Week 2:** Placebo (four 1-mL injections of placebo)

Week 4, 6, 8, 10, 12, 14: Two 1-mL injections of placebo

| Table 1 Dosing Schedule by Treatment Grot | Table 1 | Dosing Schedule by Treat | tment Group |
|---|---|---|---|
|---|---|---|---|

| Group | Baseline | Week 2 | Week 4 | Week 6 | Week 8 | Week 10 | Week 12 | Week 14 |
|---|---|---|---|---|---|---|---|---|
| 1 | 250 mg | Placebo | 125 mg | Placebo | 125 mg | Placebo | 125 mg | Placebo |
| 2 | 500 mg | Placebo | 250 mg | Placebo | 250 mg | Placebo | 250 mg | Placebo |
| 3 | 500 mg | 500 mg | 250 mg | 250 mg | 250 mg | 250 mg | 250 mg | 250 mg |
| 4 | Placebo | Placebo | Placebo | Placebo | Placebo | Placebo | Placebo | Placebo |

## 6.7 Study-Drug Administration

Study drug is to be administered to all patients in the clinic by designated and trained study personnel. Study drug should be prepared in advance and injected subcutaneously according to the following instructions:

- Remove study drug from refrigerated condition and allow to warm to room temperature for 15 minutes prior to administration. Study drug should be administered within 4 hours.
- Identify location for injections. Study drug may be injected in the abdomen, upper arm, or thigh. All injections administered at a single visit should be given in the same area, but may be split up into different areas for Week 0 and Week 2, which have 4 injections/visit. Injection sites should be ≥10 cm from one another. If possible, injections should not be administered at sites with active AD or other skin lesions.
- Inject study drug subcutaneously.
- Record location of study injections in the eCRF.
- Properly dispose of used syringe according to site requirements. Syringe box must be kept for full drug accountability.

## 6.8 Concomitant Medications and Procedures

All medications (including over-the-counter drugs, vitamins, and antacids) and over-the-counter emollient(s) taken/used at screening and throughout the study must be recorded.

The sponsor will provide the patient with an over-the-counter emollient. The patient may continue her/his current over-the-counter emollient regimen, if approved by the Investigator.

All medications and treatments taken for AD prior to screening will be recorded separately on an AD medication-history eCRF.

Patients should be instructed to consult with the Investigator prior to initiating any new medication (either self-administered non-prescription drugs or prescription therapy prescribed by another physician) while participating in the study. The Investigator is expected to examine the acceptability of all concomitant medications, topical preparations, and dietary supplements taken by patients participating in the trial.

- Medication entries should be specific to product name (if a combination drug product) and spelled correctly.
- The brand and specific product name for any over-the-counter emollient(s) should be noted and spelled correctly.
- Information on the dose, unit, frequency, route of administration, start date, discontinuation date, indication, and reason for use will be recorded.

Protocol: DRM06-AD01 A2 Page 25 Confidential

 The use of any concomitant medication must relate to an AE listed on the AE eCRF or the patient's medical history unless it is a supplement or used as preventative care.

## 6.9 Permitted and Prohibited Treatments and Procedures

The use of concomitant medications for other medical conditions (e.g., hypertension, diabetes, acute infections) is permitted during this study. Inhaled corticosteroids to control asthma are permitted.

The introduction of medications or therapies for other medical conditions known to affect AD (e.g., systemic corticosteroids, mycophenolate-mofetil, IFN-y, Janus kinase inhibitors, TCS (except when given for rescue therapy), TCI, cyclosporine, azathioprine, methotrexate, phototherapy, or photochemotherapy) are not permitted during the study and during the interval prior to entry into the study as defined in the exclusion criteria. In addition, the use of a tanning booth/parlor is not permitted during the trial.

Planned or anticipated major medication procedures or surgeries should be avoided during the trial.

## 6.10 Rescue Therapy

Patients requiring rescue therapy should consider the addition of TCS prior to considering systemic treatment. Any patient who requires TCS treatment may stay in the study and should continue the TCS for as brief a period as possible. Any patient requiring systemic therapy to treat their AD during the study will be discontinued from the study and the end of study visit assessment should be completed per Schedule of Visits and Procedures. TCS use must be recorded on the concomitant medications eCRF, indicated as "AD therapy".

## 7 STUDY PROCEDURES

The required procedures for each study visit are outlined in the study Schedule of Visits and Procedures. The timing of each study day is relative to the day of initial dosing (Day 1, Baseline).

## 7.1 Screening Visit

The purpose of the screening visit/period is to ensure that appropriate patients are entered into the study and that they remain stable during the pre-treatment period.

- Obtain written informed consent prior to performing any study procedures.
- Review Inclusion/Exclusion Criteria.
- Collect demographic information.
- Complete medical history/review of systems.
- Collect concomitant-medication and procedure/therapy information.
- Perform a complete physical examination, including height and weight.
- Measure vital signs.
- Draw blood samples for laboratory tests, including serum pregnancy test (screening visit only).
- Collect urine sample for urinalysis.
- Complete the following assessments:

- Investigator's Global Assessment (IGA)
- Eczema Area and Severity Index (EASI)
- Body Surface Area (BSA)
- Instruct the patient to apply an emollient twice daily.
- Schedule next visit.

## 7.2 Baseline Visit (Day 1)

- · Confirm emollient use.
- Re-assess and confirm patient eligibility (Inclusion/Exclusion criteria).
- Measure weight and vital signs.
- Collect concomitant medication and procedure/therapy information.
- Query for adverse events (AEs) since the last visit.
- Collect a 12-lead ECG.
- Draw blood samples for laboratory tests (hematology and chemistry)
- Draw a pre-dose blood sample for PK and anti-drug antibody (ADA) testing.
- Conduct urine for urinalysis and urine pregnancy test (WOCBP only).
- Dispense electronic tablet that will be used for home recording of pruritus NRS and sleep-loss NRS (daily), and ADIQ (weekly).
- Train patient on the use of the electronic tablet.
- Review compliance report on the electronic tablet for the assessments (pruritus NRS, sleep-loss NRS, and ADIQ) and remind patient to record daily.
- Complete the following assessments:
  - Investigator's Global Assessment (IGA)
  - Eczema Area and Severity Index (EASI)
  - Body Surface Area (BSA)
  - Patient Oriented Eczema Measure (POEM)
  - Dermatology Life Quality Index (DLQI)
  - Hospital Anxiety and Depression Scale (HADS).
- Randomize the patient.
- Administer study drug.
- Instruct the patient to apply an emollient twice daily.
- Schedule next visit.

## 7.3 Visits on Day 15, Day 29, Day 43, Day 57, Day 71, Day 85 and Day 99 (+/- 3 Day)

Confirm emollient use.

- Measure vital signs.
- Collect concomitant-medication information.
- Review and record AEs.
- Review compliance report on the electronic tablet for the daily assessments (pruritus NRS, sleep-loss NRS, and ADIQ) and remind patient to continue daily record.
- At **Day 29, 57, and 85**, draw blood samples for laboratory tests, and collect urine for urinalysis and pregnancy test (WOCBP only).
- At **Day 29, 57, and 85**, complete the following assessments:
  - Investigator's Global Assessment (IGA)
  - Eczema Area and Severity Index (EASI)
  - Body Surface Area (BSA)
- At Day 57 complete the following assessments:
  - Dermatology Life-Quality Index (DLQI)
  - Hospital Anxiety and Depression Scale (HADS).
- At Day 15, 29, 57, and 85, collect blood samples for PK (see Section 8.2.2 for instructions).
- At **Day 15 and 29**, collect a pre-dose blood sample for ADA testing (see Section 8.2.2 for instructions).
- Administer study drug.
- Remind the patient to apply an emollient twice daily.
- Remind the patient to use the tablet daily.
- Schedule next visit.

## 7.4 Visit Day 113 (Week 16) (+/- 3 Day) (End-of-Treatment/Early-Termination Visit)

Patients who discontinue the study early for any reason should have these assessments performed at their early-termination visit. The reason for early termination must be recorded in the patient's records and the eCRF.

- Confirm emollient use.
- Perform a complete physical examination, including weight.
- Measure vital signs.
- Collect concomitant medication and procedure/therapy information.
- Review and record AEs.
- Collect a 12-lead ECG.
- Draw blood samples for laboratory tests (hematology and chemistry).
- Draw a blood sample for PK and ADA testing.
- Collect urine for urinalysis and urine pregnancy test (WOCBP only).

- Review compliance report on the electronic tablet for the daily assessments (pruritus NRS, including a global impression of change for itching; sleep-loss NRS; and ADIQ).
- Collect electronic tablets and download any remaining data on device.
- Complete the following assessments:
  - Investigator's Global Assessment (IGA)
  - Eczema Area and Severity Index (EASI)
  - Body Surface Area (BSA)
  - Patient-Oriented Eczema Measure (POEM)
  - Dermatology Life Quality Index (DLQI)
  - Hospital Anxiety and Depression Scale (HADS)
  - Global Assessment of Change for AD.
- Remind the patient to apply an emollient twice daily.
- Schedule next visit.

## 7.5 Follow-Up Visit Day 141 (Week 20) (+/- 7 Days)

- Measure vital signs.
- Collect concomitant medication and procedure/therapy information.
- Review and record AEs.
- Complete the following assessments:
  - Investigator's Global Assessment (IGA)
  - Eczema Area and Severity Index (EASI)
- Remind the patient to apply an emollient twice daily
- Schedule next visit.

## 7.6 Follow-Up Visit Day 169 (Week 24) (+/- 7 Days)

- Measure vital signs.
- Collect concomitant medication and procedure/therapy information.
- Review and record AEs.
- Draw blood samples for laboratory tests (hematology and chemistry)
- Draw blood sample for PK and ADA testing.
- Collect urine for urinalysis and urine pregnancy test (WOCBP only).
- Complete the following assessments:
  - Investigator's Global Assessment (IGA)
  - Body Surface Area (BSA).
  - Eczema Area and Severity Index (EASI)

- Remind the patient to apply an emollient twice daily
- Add reminder to schedule a FU visit phone call.

## 7.7 Follow-Up Visit Phone Call, Day 225 (Week 32) (+/- 7 Days)

Review and record AEs.

#### 7.8 Unscheduled Visits

If an unscheduled visit is necessary, the following assessments should be included in the visit along with any assessments that are the reason for the visit (e.g., blood draw for a repeat of abnormal lab values):

- Measure vital signs.
- Collect concomitant medication and procedure/therapy information.
- Review and record AEs.

#### 8 DETAILS OF ASSESSMENTS

## 8.1 Screening Assessments

## 8.1.1 Demographics

At the screening visit, demographic information including age, gender, race and ethnicity will be collected and recorded in the eCRF for each patient.

## 8.1.2 Medical History

A complete medical history will be collected as part of the screening assessment and include all clinically relevant past or coexisting medical conditions or surgeries. Extensive information on the patient's atopic dermatitis, asthma, and allergies will be collected as part of the medical history. The medical history will be updated prior to treatment on Baseline/Day 1 should new findings be present since the screening visit. Findings will be recorded in the eCRF.

#### 8.1.3 Disease Specific Information

Information on the patient's atopic dermatitis will be collected as part of the screening assessment and include the date of onset of atopic dermatitis, anatomical areas affected by atopic dermatitis, and past treatments for atopic dermatitis. Information will be recorded in the eCRF.

## 8.2 Assessment of Efficacy

#### 8.2.1 AD Assessments

Each patient's AD will be assessed as specified in the Schedule of Visits and Procedures. Whenever possible, the same assessor should perform all assessments on a given patient. Individuals will be trained and certified by the Sponsor prior to conducting any assessments.

#### 8.2.1.1 Investigator Global Assessment (IGA)

The IGA (Appendix 3) is an instrument used to globally rate the severity of the patient's AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). The IGA must be conducted prior to conducting the EASI assessment.

A grade of 0 to 4 will be assessed by the Investigator or designee. Assessors must be trained and certified by the Sponsor prior to conducting this assessment. Assessments will be recorded in the eCRF.

## 8.2.1.2 Eczema Area and Severity Index (EASI)

The EASI (Appendix 4) is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with the higher values indicating more severe and or extensive disease. A grade of 0 to 72 will be assessed by the Investigator or designee.

Assessors must be trained and certified by the Sponsor prior to conducting this assessment. Assessments will be recorded in the eCRF.

## 8.2.1.3 Body Surface Area (BSA)

The BSA (Appendix 5) assessment estimates the extent of disease or skin involvement with respect to AD and is expressed as a percentage of total body surface. BSA will be determined by the Investigator or designee using the patient palm = 1% rule.

Assessments will be recorded in the eCRF. Assessors must be trained and certified by the Sponsor prior to conducting this assessment.

#### 8.2.1.4 **Pruritus**

Pruritus will be assessed by the patient using a Pruritus Numeric Rating Scale (NRS) (Appendix 6). The Pruritus NRS is an 11-point scale used by patients to assess their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable". At Week 16, a global impression of change for itching question will be requested.

Assessments will be recorded daily by the patient using an electronic diary and transferred into the clinical database.

## 8.2.1.5 Sleep-Loss

Quality of sleep will be assessed by the patient using a sleep-loss question (Appendix 7) over the past 24 hours.

Assessments will be recorded daily by the patient using an electronic diary and transferred into the clinical database.

## 8.2.1.6 Atopic Dermatitis Impact Questionnaire (ADIQ)

The ADIQ (Appendix 8) is a 17-item questionnaire used to assess the patients' AD-specific health-related QoL. The questionnaire assesses AD's impact on emotions, energy, activities of daily living, and social activities. The ADIQ has a recall specification of 7 days.

Assessments will be recorded by the patient using an electronic diary and transferred into the clinical database.

## 8.2.1.7 Patient Oriented Eczema Measure (POEM)

The POEM (Appendix 9) is a 7-item questionnaire used by the patient to assess the severity of the patient's eczema over the last week. All seven answers carry equal weight and are scored as: No days=0; 1– 2 days =1; 3–4 days=2; 5–6 days=3; everyday=4.

The POEM is completed by the patient in the clinic. Assessments will be recorded in the eCRF.

## 8.2.1.8 Dermatology Life Quality Index (DLQI)

The DLQI (Appendix 10) is a 10-question instrument used to measure the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, over the previous week.

Questions are scored from 0 to 3, giving a possible total score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).

The DLQI is completed by the patient in the study clinic. Assessments will be recorded in the eCRF.

## 8.2.1.9 Hospital Anxiety and Depression Scale (HADS)

The HADS (Appendix 11) assesses anxiety and depression in a non-psychiatric population. The HADS has two subscales (depression and anxiety), both with 7 questions.

Responses are based on the relative frequency of symptoms over the past week, using a four-point scale ranging from 0 (not at all) to 3 (very often indeed).

HADS is completed by the patient in the clinic. Assessments will be recorded in the eCRF.

## 8.2.1.10 Global Assessment of Change-AD

The Global Assessment of Change for AD (Appendix 12) will be one question asked at Week 16 and the Early-Termination visit. The value of the question is to capture the patient's impression of overall change in their AD.

This will be completed by the patient in the clinic. Assessments will be recorded in the eCRF

## 8.2.2 PK and ADA Sampling

Serum PK and ADA samples on Day 1, 15, 29, 57 (PK only), 85 (PK only), 113, and 169 will be taken predose. PK and ADA samples will be collected from all patients including those assigned to the placebo group to maintain the blinding of the treatment assignment. Positive ADA results will be further evaluated for antidrug antibodies. The procedural instructions will be provided in a separate PK and Serum Antibody Sampling manual.

#### 9 ASSESSMENT OF SAFETY

## 9.1 Assessment of Safety

## 9.1.1 Physical Examination

A complete physical examination will be conducted at screening and cover general appearance, dermatological, head, ears, eyes, nose, throat, respiratory, cardiovascular, abdominal, neurological, musculoskeletal, and lymphatic body systems. Height and weight will be recorded as part of the screening physical exam and only the patient's weight will be recorded with the Baseline and the week 16 physical examination. Findings will be recorded in the eCRF.

At subsequent study visits, a symptom-directed physical examination may be conducted.

## 9.1.2 Vital Signs

Vital signs, including body temperature, respiratory rate (breath per minute), pulse (beats per minute), and blood pressure (mmHg), will be obtained with the patient in the seated position,

after sitting for at least 5 minutes. Any abnormal findings which are new or worsened in severity and clinically significant, in the opinion of the Investigator, will be recorded as an AE. Vital sign measurements will be recorded in the eCRF.

#### 9.1.3 ECGs

12-lead ECG measurements will be obtained in all patients. The patient should rest quietly for at least 5 minutes in a supine position prior to ECG collection. The ECG should be obtained either prior to the time of blood collection, or at least 15 minutes afterwards. The medical monitor may be consulted if needed for interpretation of ECGs.

All study sites will be supplied with standardized, validated, digital, 12-lead ECG machine (12-lead at 25 mm/sec reporting rhythm, ventricular rate, the RR interval, the PR interval, QRS duration, QT and QTcF intervals) capable of recording, storing, printing, and producing high resolution 12-lead ECG data. Study sites will be trained on the use of the equipment prior to study start.

Machine-read ECG recordings will be collected and analyzed centrally. Data will be transferred electronically to the database.

#### 9.1.4 Laboratory Evaluations

Laboratory tests will be analyzed using a central laboratory and include hematology with differential, serology, a standard chemistry panel (including liver-function tests), total cholesterol, standard urine testing, and urine pregnancy test for women of child-bearing potential (WOCBP). Blood and urine will be collected from each patient as specified in the Schedule of Visits and Procedures or as clinically indicated. Laboratory samples are to be shipped on the same day as collected. Laboratory test results will be provided to the sites through a web-based reporting system. Alert values will be emailed to the site. Laboratory data will be transferred to the clinical database from the central laboratory database.

Screening laboratory test results must be reviewed by the Investigator prior to patient enrollment. Patients will fail screening for clinically significant laboratory values. However, at the discretion of the Investigator, screening laboratory tests may be repeated one time to confirm out-of-range results or clinical significance. Specific laboratory tests are listed in Table 2.

The central laboratory should be used for all laboratory testing required for a patient during study participation, including laboratory testing needed for unscheduled visits. Clinically significant laboratory results must be entered as a diagnosis on the AE eCRF rather than as an individual test result. Patients with clinically significant laboratory test results will be evaluated, treated and followed at the discretion of the Investigator until the value returns to clinically acceptable levels.

Throughout the study, all laboratory results should be reviewed and signed by the Investigator within 48 hours of receipt of the report (whenever possible).

**Table 2** Laboratory Parameters

| Hematology | Chemistry | Urine |
|---|---|---|
| Hematocrit (HCT) | Sodium | • pH |
| Hemoglobin (HGB) | Potassium | Specific gravity, protein |
| Red blood cells (RBC) | Chloride Calcium | Glucose |
| White blood cells (WBC) | Phosphorus | Ketones |
| Mean corpuscular | Bicarbonate | Bilirubin |
| hemoglobin (MCH) | Uric Acid | Blood |
| MCH concentration | Blood urea nitrogen (BUN) | Nitrite |
| (MCHC) | Creatinine | Urobilinogen |
| Mean corpuscular volume (MCV) | Total Protein | Leukocyte esterase |
| RBC morphology | Albumin | At all visits except screening |
| Platelet count | Aspartate aminotransferase | (WOCBP only): Urine beta human chorionic gonadotropin (β-hCG) |
| Neutrophils | (AST) | |
| Lymphocytes | Alanine aminotransferase (ALT) | |
| Monocytes | Lactic dehydrogenase (LDH) | |
| Eosinophils | Gamma-glutamyl | |
| Basophils | transpeptidase (GGT) | |
| Screening only: | Alkaline phosphatase | |
| HIV Antibody (HIV Ab) | Bilirubin (total and direct) | |
| Hepatitis B Antibody | Total cholesterol | |
| (HBcAb) Hepatitis B<br>Antigen (HBsAg) | Non-fasting glucose | |
| Hepatitis C Antibody (Hep C Ab) | For all female patients (WOCBP) at Screening: | |
| (Hep C Ab) | Serum beta human chorionic gonadotropin (β-hCG) | |

## 9.1.5 Adverse Events (AEs)

An AE is defined as any untoward medical occurrence associated with the use of a study drug in humans, whether considered drug related. An AE can, therefore, be any unfavorable and unintended sign (including clinically significant abnormal laboratory finding), symptom or disease temporally associated with the use of the study drug, whether related to the investigational product.

AEs will be monitored throughout the study. Patients will be instructed to inform the Investigator and/or study staff of any AEs. At each visit, patients will be asked about AEs in a non-specific manner using open-ended questions so as not to bias the response (e.g., How have you been since the last visit?). Specific inquiry regarding reported AEs will be conducted when applicable. All AEs will be documented and recorded in the patient's eCRF.

Any patient who has an AE (serious or non-serious) will be evaluated by the Investigator and treated and followed until the symptom(s) return to normal or to clinically acceptable levels, as judged by the Investigator. A physician, either at clinical site, or at a nearby hospital emergency room, will administer treatment for any serious AEs (SAEs), if necessary. When appropriate, medical tests and examinations will be performed to document resolution of event(s).

## **9.1.5.1** Reporting

Only AEs that occur during or following study treatment with the study drug will be reported in the AE section of the eCRF. Events recorded prior to study treatment with the drug will be reported in the Medical History section of the eCRF. All AEs occurring during the study will be individually recorded in the eCRF. Any condition present prior to administration of study drug and that worsens after administration of study drug should be reported as an AE. Information regarding the onset, duration, severity, action taken, outcome, and relationship to study drug will be recorded.

New or worsening abnormal laboratory values and/or vital signs are to be recorded as AEs if they are considered to be of clinical significance by the Investigator or meet the criteria of an SAE as described in Section 9.1.6. Unless a diagnosis is available, signs and symptoms must be reported as individual AEs in the eCRF; a diagnosis is preferred.

The severity of an AE will be designated as mild, moderate or severe. The term "severe" is used to describe the intensity of an AE; the event itself, however, may be of relatively minor clinical significance (e.g., 'severe' upper respiratory infection). Severity is not the same as "serious". Seriousness of AEs is based on the outcome/action of an AE. (See Section 9.1.6.)

The relationship of the AE to the study treatment should be determined by the Investigator and will be based on the following two definitions:

**Not related**: The AE is judged to not be associated with the study drug, and is attributable to another cause.

**Related:** A causal relationship between the AE and the study drug is a reasonable possibility, i.e., there is evidence (e.g., dechallenge/rechallenge) or other clinical arguments to suggest a causal relationship between the AE and study treatment.

## 9.1.6 Serious Adverse Events (SAEs)

An SAE is defined as any untoward medical occurrence that,

- Results in death
- Is in the opinion of the Investigator immediately life threatening (i.e., the patient is at immediate risk of death; it does not include a reaction that, had it occurred in a more severe form, might have caused death)
- Requires inpatient hospitalization or results in prolongation of an existing hospitalization
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly or birth defect
- Is an important medical event that may not be immediately life-threatening, result in death, or require hospitalization, but based on appropriate medical judgment, it jeopardizes the patient, or may require medical or surgical intervention to prevent one of the outcomes listed.

The Investigator should institute any clinically necessary supplementary investigation of SAE information. In the case of patient death, any post-mortem findings/reports will be requested.
### 9.1.6.1 Reporting of SAEs

All SAEs, as defined in Section 9.1.6, regardless of causal relationship, must be reported to the Sponsor or designee within 24 hours of the Investigator becoming aware of the event. As soon as the Investigator becomes aware of an AE that meets the criteria for an SAE, the SAE should be documented to the extent that information is available.

SAEs will be recorded from the time of informed consent/assent until the end of the study. If, in the opinion of the Investigator, an SAE occurring outside the specified time window (i.e., following patient completion or terminations of the study) is deemed to be drug-related, the event should be reported with 24 hours.

SAEs must be recorded on an SAE form. The minimum information required for SAE reporting includes the identity of the PI, site number, patient number, event description, SAE term(s), reason why the event is considered serious (i.e., the seriousness criteria), and PI's assessment of the relationship of the event to study drug. Additional SAE information including medications or other therapeutic measures used to treat the event, and the outcome/resolution of the event should also be recorded on the SAE form.

In all cases, the Investigator should continue to monitor the clinical situation and report all material facts relating to the progression or outcome of the SAE. The Investigator may be required to provide supplementary information as requested by the Sponsor or its designee.

When reporting SAEs, the following additional points should be considered:

- Although signs, symptoms, and tests that support the diagnosis of an SAE should be provided, the Investigator should report the diagnosis or syndrome as the SAE term.
- Death should not be reported as an SAE, but as an outcome of a specific SAE (unless
  the event preceding the death is unknown). If an autopsy was performed, the autopsy
  report should be provided.

Although most hospitalizations necessitate reporting of an SAE, some hospitalizations do not:

- Hospitalization for elective or previously scheduled surgery, or for a procedure for a preexisting condition that has not worsened after administration of study drug (e.g., a
  previously scheduled ventral hernia repair). SAEs must, however, be reported for any
  surgical or procedural complication that lead to prolongation of the hospitalization.
- Events that result in hospital stays for observation of <24 hours and that do not require a therapeutic intervention/treatment (e.g., an emergency room visit for hematuria that results in a diagnosis of cystitis and discharge to home on oral antibiotics).

The Sponsor will process and evaluate all SAEs as soon as the reports are received. For each SAE received, the Sponsor will determine whether the criteria for expedited reporting to relevant regulatory authorities have been met.

The Sponsor will assess the likelihood that each SAE is related to study treatment, with the current Investigator's Brochure used as the reference document to assess expectedness of the event to study drug.

#### 9.1.7 Adverse Events of Special Interest (AESI)

AESIs in this study include:

- Anaphylactic reactions or acute allergic reactions that require immediate treatment
- Malignancies (excluding non-melanoma skin cancers).

All AESIs must be reported to the sponsor and designee within 24 hours of identification.

### 9.1.8 Pregnancy

In the instance that a patient becomes pregnant during participation in the study, the patient must be withdrawn from study drug but may continue study participation. The Investigator must perform medical assessments as clinically indicated and continue to follow the patient for ≥4 weeks after delivery, at a minimum. Details for both the mother and baby must be obtained.

Although pregnancy is not itself an AE or SAE, maternal/fetal complications or abnormalities will be recorded as AEs or SAEs, as appropriate.

The Investigator must complete a study-specific Pregnancy Form upon confirmation of a pregnancy. Pregnancy reporting forms will be provided to the site.

# 10 STUDY DISCONTINUATIONS

### 10.1 Study Termination

The Sponsor has the right to terminate or to stop the study at any time. Should the study be terminated, the decision and reason will be communicated in writing by the Sponsor to the Investigator and request that all patients be discontinued. Should this be necessary, patients should be scheduled for an Early-termination visit (Section 7.4).

The entire study will be stopped if:

- Evidence has emerged that, in the collective opinion of the Investigators at each site with the concurrence of the Sponsor, or the sole opinion of the Sponsor, continuation of the study is unnecessary or unethical
- The stated objectives of the study are achieved
- The Sponsor discontinues the development of the study drug

If the study is terminated by the Sponsor, all data available for the patient at the time of discontinuation must be recorded in the patient's records and the eCRF.

#### 10.2 Early Termination of Study Patients

The Investigator will make every reasonable effort to keep each patient in the study. However, patients may terminate or be terminated early from the study for the following reasons:

- Voluntarily withdrawal of consent to participate in the study participation, at any time
- Adverse event, laboratory abnormality or inter-current illness which, in the opinion of the Investigator, indicates that continued treatment and/or participation in the study is not in the best interest of the patient
- Serious protocol violation, persistent non-compliance or requirement for medication or procedure prohibited by the protocol
- Lost to follow-up

Patients who are terminated early from study will have an Early-Termination visit scheduled (Section 7.4) as soon as possible. All information, including the reason for early discontinuation will be recorded in the patient's study records and in the eCRF.

Before a patient can be terminated early due to loss of follow-up, the Investigator must show documented attempts to contact the patient regarding study participation on two separate occasions (telephone contact) followed by a certified letter of contact.

Prior to discontinuing a patient from study participation, the Investigator will discuss his/her intentions with the Sponsor Medical Monitor or designee.

## 10.3 Study-Drug Discontinuation

Study drug must be discontinued for patients who experience the following:

- Inter-current illness that would, in the judgment of the Investigator, affect assessments of clinical status to a significant degree
- Treatment related AEs that are clinically significant, deemed persistent, in the judgment of the Investigator
- Unacceptable toxicity
- Pregnancy

Patients who discontinue study drug permanently during study participation must be scheduled for an Early-termination visit (Section 7.4).

#### 11 STATISTICAL CONSIDERATIONS

### 11.1 General Statistical Methodology

All statistical processing will be performed using SAS<sup>®</sup> unless otherwise stated. No interim analyses are planned.

Except where noted, all statistical tests will be two-sided and will be performed at the 0.05 level of significance. The inclusion of p-values in the efficacy analyses is to assist in characterizing the therapeutic efficacy of the active medication. No adjustments will be made for multiple comparisons for the efficacy analyses. The primary analysis will be performed when all patients have completed the treatment phase at Week 16. The final time-course data analysis will be performed when all patients have finished Week 32.

Descriptive statistics will be used to provide an overview of the efficacy and safety results. For categorical parameters, the number and percentage of patients in each category will be presented. The denominator for percentage will be based on the number of patients appropriate for the analysis. For continuous parameters, descriptive statistics will include the number of patients (n), mean, standard deviation (SD), median, and range. Appropriate inferential statistics will be used for the primary and secondary efficacy variables.

For the primary efficacy variable, the primary method of handling missing efficacy data will be the method of MCMC multiple imputation. This method does not rely on the assumption of data missing at random. Additionally, imputation will be conducted within each treatment group independently so the pattern of missing observations in one treatment group cannot influence missing value estimations in another.

For binary responses related to EASI and IGA, the binary response variables will be calculated based on the multiply imputed datasets that have been created. Because the MCMC algorithm is based on the multivariate normal model, imputed values for IGA will not generally be one of the discrete values used in IGA scoring (0, 1, 2, 3, or 4). Therefore, to derive the binary IGA response variable, standard rounding rules will be applied to the imputed values. For example, if a patient has a IGA score imputed as 1.4 (and assuming a Baseline IGA score of 3), the imputed value would be rounded down to 1, and the minimum change from Baseline of 2 would have been met. This patient would be considered a responder.

DRM06-AD01-A2

For derivation of EASI75 response, no rounding will be performed. The imputed Week 16 EASI value will be compared directly to the observed Baseline EASI value to determine whether a reduction of at least 75% was achieved.

For the EASI assessment, a total of 4 seeds are required to impute the EASI score for the four treatment groups. Those 4 random seeds have been pre-specified by using a random number generator:

```
Lebrikizumab, 125 mg every 4 weeks: seed = 1083679005
Lebrikizumab, 250 mg every 4 weeks: seed = 1346533179
Lebrikizumab, 250 mg every 2 weeks: seed = 297484487
Placebo every 2 weeks: seed = 424603513
```

For the IGA assessment, a total of 4 seeds are required to impute the IGA score for the four treatment groups. Those 4 random seeds have been pre-specified by using a random number generator:

```
Lebrikizumab, 125 mg every 4 weeks: seed = 1975600090
Lebrikizumab, 250 mg every 4 weeks: seed = 1260832817
Lebrikizumab, 250 mg every 2 weeks: seed = 2036512379
Placebo every 2 weeks: seed = 202520365
```

Sensitivity analyses on some of the secondary efficacy variables will be performed as follows:

- Non-response imputation (NRI) will be used to impute missing values. Specifically, any patient with a missing IGA (or EASI75) value at Week 16 will be treated as a non-responder for analysis purposes.
- Demographic data will be summarized by treatment group using descriptive statistics. Patients' baseline characteristics related to efficacy analyses will be compared with descriptive statistics among treatment groups to determine whether the results are directly comparable.
- The number of patients in each analysis set will be summarized. Reasons for study withdrawal during the blinded study will be summarized using frequencies and percentages by treatment group.

A statistical analysis plan (SAP) describing all statistical analyses will be provided as a separate document. The SAP will be finalized prior to unblinding of the treatment groups.

### 11.2 Populations Analyzed

Patients will be randomized in a 3:3:3:2 ratio to each treatment group. There will be approximately 75 patients for groups with study drug, and 50 patients for the placebo group.

Efficacy analyses will be performed using the modified intent-to-treat (mITT) population and the per-protocol (PP) population. The mITT population will include all patients who were randomized and received study drug. The PP population will include all patients in the safety population who completed the Week 16 evaluation without any significant protocol violations (i.e., any patient or Investigator activity that could have possibly interfered with the therapeutic administration of the treatment or the precise evaluation of treatment efficacy).

Safety analyses will be performed using the safety population. All patients who are randomized and receive ≥1 dose of study drug will be included in the safety population.

# 11.3 Primary Efficacy

The following primary endpoint will be analyzed:

Percent change in Eczema Area and Severity Index (EASI) from Baseline to Week 16.

# 11.4 Secondary Efficacy

The following secondary endpoints will be analyzed:

- Proportion of patients with a 75% improvement from Baseline in EASI (EASI75) at Week 16.
- Proportion of patient with an IGA score of 0 (clear) or 1 (almost clear) and a reduction
   ≥2 points from Baseline to Week 16.
- Proportion of patients with EASI <7 at Week 16.</li>
- Proportion of patients achieving EASI50 and EASI90 at Week 16.
- Percent change in sleep-loss numerical rating scale (NRS) score from Baseline to Week 16.
- Percent change in pruritus numerical rating scale (NRS) score from Baseline to Week 16.
- Proportion of patients with pruritus NRS change of ≥3 from Baseline to Week 16.
- Proportion of patients with pruritus NRS change of ≥4 from Baseline to Week 16.
- Change in Body Surface Area (BSA) involved with AD from Baseline to Week 16.

## 11.5 PK Analysis

Plasma concentration data will be tabulated and summarized (geometric mean, arithmetic mean, minimum, maximum, SD, and % coefficient of variation) by treatment group for each visit at which samples were taken.

The planned PK analysis will be included in a separate Pharmacokinetic Analysis Plan.

#### 11.6 Exposure and Compliance

The extent of exposure to study drug in each treatment group will be summarized by total number of days of exposure, total number of applications, number of missed applications, and number and percentage of patients who are compliant. An application is considered the full set of injections (either 2 or 4 depending on visit) specified by the protocol.

A patient will be considered compliant with the dosing regimen if the patient received ≥75% of the expected number of applications while enrolled in the study.

#### 11.7 Adverse Events

All AEs occurring during the study will be recorded and coded using the MedDRA dictionary. Treatment-emergent AEs (TEAEs) are defined as AEs with an onset date on or after the date of the first application. TEAEs will be summarized by treatment group, including the number of patients reporting an event, system organ class, preferred term, severity, relationship to study drug, and seriousness for the safety population. All serious AEs as well as AEs that led to study discontinuation will be listed by patient.

Three sets of AE tabulations are anticipated, one for the treatment period, one for the post-treatment (follow-up) period, and one for the combined treatment and post treatment period. The denominator used for the treatment period will correspond to the number of patients in the safety population. Data will also be corrected for exposure and reported per 100 patient-years.

# 11.8 Other Safety Data

Laboratory data will be presented in a by patient listing. Any clinically significant laboratory abnormalities will be captured as AEs. Changes from Baseline in safety laboratory values will be summarized by treatment group at each follow-up evaluation during the treatment period using descriptive statistics or frequency tables as applicable. Tables and listings will be in SAS format. Additionally, changes from Baseline in safety laboratory values will be summarized using shift tables according to normal ranges.

ECGs and vital signs will be presented by treatment group as absolute values and changes from Baseline using descriptive statistics.

Medical histories will be coded using the MedDRA dictionary and presented in a by-patient listing. Concomitant medications will be coded using the WHO-Drug dictionary. Concomitant medications will be summarized by treatment, drug class, and preferred term. Physical examination data will be presented in a by-patient listing.

## 11.9 Sample-Size Determination

The sample size for this study was based mainly on clinical considerations.

#### 12 ADMINISTRATION

### 12.1 Compliance with the Protocol

The study shall be conducted as described in this protocol. All revisions to the protocol must be prepared by the Sponsor. The Investigator will not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion from the IRB/IEC of an Amendment, except where necessary to eliminate an immediate hazard(s) to study patients. Any significant deviation must be documented and submitted to the: IRB/IEC; the Sponsor or designee; and, if required, Regulatory Authority(ies). Documentation of approval signed by the chairperson or designee of the IRB(s)/EC(s) must be sent to the Sponsor and/or designee.

## 12.2 Informed Consent Procedures

The Informed Consent Form (ICF) will include all elements required by ICH/GCP and applicable regulatory requirements, and will adhere to GCP and to the ethical principles that have their origin in the Declaration of Helsinki. The consent form will also include a statement that the Sponsor and regulatory authorities have direct access to patient records.

Prior to the beginning of the study, the Investigator will have the IRB/IEC's written opinion (approval/favorable) of the written informed consent form and any other information to be provided to the patients.

The Investigator must provide the patient or legally acceptable representative with a copy of the consent form and written information about the study in the language in which the patient is most proficient. The language must be non-technical and easily understood. The Investigator should allow time necessary for patient or patient's legally acceptable representative to inquire about the details of the study, then informed consent must be signed and personally dated by the patient or the patient's legally acceptable representative, by the Investigator and by the

person who conducted the informed consent discussion. The patient or legally acceptable representative should receive a copy of the signed informed consent and any other written information provided to study patients prior to patient's participation in the study.

The informed consent and any other information provided to patients or the patient's legally acceptable representative, should be revised whenever important new information becomes available that is relevant to the patient's consent, and should receive IRB/IEC approval/favorable opinion prior to use. The Investigator, or a person designated by the Investigator should fully inform the patient or the patient's legally acceptable representative of all pertinent aspects of the study and of any new information relevant to the patient's willingness to continue participation in the study. This communication to the patient should be documented in the source note.

During a patient's participation in the study, any updates to the consent form or to the written information will be provided to the patient in writing.

### 12.3 Study Documentation and the eCRF

This protocol is to be signed by the investigator responsible for the conduct of this study at the study site. A copy of the signed protocol signature page is to be provided to the Sponsor and retained in the study site's Regulatory Binder.

The Investigator is responsible for ensuring that all study data is accurately recorded on the eCRFs or other study data collection tools. All eCRF entries must be supported by the patient's medical records or source notes. The Investigator must ensure that study observations and findings are legible and recorded accurately and completely.

Original reports, traces and films must be reviewed, signed and dated, and retained by the Investigator for future reference.

The Investigator is expected to promptly review all study data recorded in the patient's source records. Completed eCRFs must be promptly reviewed, signed, and dated by the Investigator or Sub-Investigator at the end of the study. Corrections to data entered into the eCRF will be handled through an electronic query. Corrections to patients' medical or source records should be legible, initialed and dated. At the end of the study, an electronic copy of the investigator's eCRFs will be provided to the Investigator. The Investigator is to retain this data. The Investigator will maintain a signature sheet to document signatures and initials of all persons authorized to make entries and/or corrections on eCRFs. Refer to Section 12.5 regarding retention requirements.

An Investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation for each patient treated with the study drug or entered as a control in the investigation. Data reported on the eCRFs that are derived from source documents must be consistent with the source documents or the discrepancies must be explained.

#### 12.4 Study Monitoring

The Sponsor or designee will be responsible for the monitoring of the study. Study monitors will contact and visit the Investigators at regular intervals throughout the study to verify adherence to the protocol, and assess the completeness, consistency, and accuracy of the data by comparing patients' medical records with entries in the eCRF.

The study monitor must be allowed access to laboratory test reports and other patient records needed to verify the entries on the eCRF, provided patient confidentiality is maintained in accordance with local requirements. These records, and other relevant data, may also be

reviewed by appropriate qualified personnel independent from the Sponsor or designee, who is appointed to audit the study. Patient confidentiality will be maintained at all times.

By agreeing to participate in this research study, the Investigators agree to co-operate with the study monitor to ensure that any problems detected during the monitoring visits are promptly resolved.

# 12.5 Retention of Study Documentation

The Investigator must retain study drug disposition records, copies of CRFs and all study-related source documents for the maximum period required by applicable regulations and guidelines, or Institution procedures, or for the period specified by the Sponsor, whichever is longer. The Investigator must contact the Sponsor prior to destroying any records associated with the study.

If the Investigator withdraws from the study (e.g., relocation, retirement), the records shall be transferred to a mutually agreed upon designee (e.g., another Investigator, IRB). Notice of such transfer will be given in writing to the Sponsor or designee.

If the Investigator cannot guarantee this archiving requirement for any or all the documents at the investigational site, arrangements must be made between the Investigator and the Sponsor to store these in a secure archive facility outside the site so they can be returned to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the patient, appropriate copies should be made for storage outside of the site.

## 12.6 Acronyms

The acronyms listed below are a non-exhaustive list of those commonly used in Dermira study documents. Not all acronyms listed below are used within this document.

| Acronym | Term |
|---------|----------------------------------------|
| ADIQ | Atopic dermatitis impact questionnaire |
| AE | Adverse event(s) |
| ALT | Alanine amino-transferase |
| ASIQ | AD-specific health-related QoL |
| AST | Aspartate amino-transferase |
| AD | Atopic dermatitis |
| BP | blood pressure |
| BUN | Blood urea nitrogen |
| С | Celsius |
| CFR | Code of federal regulations |
| eCRF | Electronic case report form |
| CRO | Clinical research organization |
| EASI | Eczema area of severity index |
| ET | Early termination |
| F | Fahrenheit |
| FDA | Food and Drug Administration |
| GCP | Good clinical practice |

| Acronym | Term |
|---------|----------------------------------------------|
| GGT | Gamma-glutamyl transferase |
| GLP | Good laboratory practice |
| HCT | Hematocrit |
| HGB | Hemoglobin |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent ethics committee |
| IRB | Institutional review board |
| ITT | Intent-to-treat |
| IUD | Intrauterine device |
| IV | Intravenous |
| IWRS | Interactive web response system |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PDK | phosphoinositide-dependent kinase |
| PK | Pharmacokinetics |
| PP | Per protocol |
| QoL | Quality of life |
| Q4W | Every 4 weeks |
| RBC | Red blood cells |
| SAE | Serious adverse event(s) |
| SC | Subcutaneous |
| SCORAD | Severity scoring of atopic dermatitis |
| SOC | System organ class |
| TCS | Topical corticosteroids |
| TCI | Topical calcineurin inhibitors |
| Th-2 | T-helper type 2 |
| TEAE | Treatment-emergent adverse events |
| US | United States |
| VAS | Visual analog scale |
| WBC | White blood cells |
| WHO | World Health Organization |
| WOCBP | Women of childbearing potential |

#### 13 REFERENCES

- Gittler, JK, Shemer A, Suarez-Farinas M, et al. 2012. Progressive activation of T(H)2/T(H)22 cytokines and selective epidermal proteins characterizes acute and chronic atopic dermatitis. J Allergy Clin Immunol. 130:1344-54.
- 2. Bieber, T. 2010. Atopic dermatitis. Ann Dermatol. 22:125-37.
- 3. Bieber, T, Novak N. 2009. Pathogenesis of atopic dermatitis: new developments. Current allergy and asthma reports. 9:291-4.
- 4. Williams, H, Stewart A, von Mutius E, et al. 2008. Is eczema really on the increase worldwide? J Allergy Clin Immunol. 121:947-54 e15.
- 5. Asher, MI, Montefort S, Bjorksten B, et al. 2006. Worldwide time trends in the prevalence of symptoms of asthma, allergic rhinoconjunctivitis, and eczema in childhood: ISAAC Phases One and Three repeat multicountry cross-sectional surveys. Lancet. 368:733-43.
- 6. Shaw, TE, Currie GP, Koudelka CW, et al. 2011. Eczema prevalence in the United States: data from the 2003 National Survey of Children's Health. J Invest Dermatol. 131:67-73.
- 7. Hanifin, JM, Reed ML, Eczema P, et al. 2007. A population-based survey of eczema prevalence in the United States. Dermatitis. 18:82-91.
- 8. Emerson, RM, Williams HC, Allen BR. 1998. Severity distribution of atopic dermatitis in the community and its relationship to secondary referral. The British journal of dermatology. 139:73-6.
- Silverberg, JI, Simpson EL. 2013. Association between severe eczema in children and multiple comorbid conditions and increased healthcare utilization. Pediatr Allergy Immunol. 24:476-86.
- 10. Zuberbier, T, Orlow SJ, Paller AS, et al. 2006. Patient perspectives on the management of atopic dermatitis. J Allergy Clin Immunol. 118:226-32.
- 11. Kiebert, G, Sorensen SV, Revicki D, et al. 2002. Atopic dermatitis is associated with a decrement in health-related quality of life. International journal of dermatology. 41:151-8.
- 12. Ring, J, Alomar A, Bieber T, et al. 2012. Guidelines for treatment of atopic eczema (atopic dermatitis) Part II. Journal of the European Academy of Dermatology and Venereology: JEADV. 26:1176-93.
- 13. Schneider, L, Tilles S, Lio P, et al. 2013. Atopic dermatitis: a practice parameter update 2012. J Allergy Clin Immunol. 131:295-9 e1-27.
- 14. He, JQ, Chan-Yeung M, Becker AB, et al. 2003. Genetic variants of the IL13 and IL4 genes and atopic diseases in at-risk children. Genes Immun. 4:385-9.
- 15. Hummelshoj, T, Bodtger U, Datta P, et al. 2003. Association between an interleukin-13 promoter polymorphism and atopy. Eur J Immunogenet. 30:355-9.
- Novak, N, Kruse S, Kraft S, et al. 2002. Dichotomic nature of atopic dermatitis reflected by combined analysis of monocyte immunophenotyping and single nucleotide polymorphisms of the interleukin-4/interleukin-13 receptor gene: the dichotomy of extrinsic and intrinsic atopic dermatitis. J Invest Dermatol. 119:870-5.
- 17. Howell, MD, Kim BE, Gao P, et al. 2009. Cytokine modulation of atopic dermatitis filaggrin skin expression. J Allergy Clin Immunol. 124:R7-R12.
- 18. Purwar, R, Werfel T, Wittmann M. 2006. IL-13-stimulated human keratinocytes preferentially attract CD4+CCR4+ T cells: possible role in atopic dermatitis. J Invest Dermatol. 126:1043-51.

- 19. Esche, C, de Benedetto A, Beck LA. 2004. Keratinocytes in atopic dermatitis: inflammatory signals. Current allergy and asthma reports. 4:276-84.
- 20. Kim, BE, Leung DY, Boguniewicz M, et al. 2008. Loricrin and involucrin expression is down-regulated by Th2 cytokines through STAT-6. Clin Immunol. 126:332-7.
- 21. Bhogal, RK, Bona CA. 2008. Regulatory effect of extracellular signal-regulated kinases (ERK) on type I collagen synthesis in human dermal fibroblasts stimulated by IL-4 and IL-13. Int Rev Immunol. 27:472-96.
- 22. Kim, ST, Lee KM, Park HJ, et al. 2009. Topical delivery of interleukin-13 antisense oligonucleotides with cationic elastic liposome for the treatment of atopic dermatitis. J Gene Med. 11:26-37.
- 23. Akdis, M, Akdis CA, Weigl L, et al. 1997. Skin-homing, CLA+ memory T cells are activated in atopic dermatitis and regulate IgE by an IL-13-dominated cytokine pattern: IgG4 counter-regulation by CLA- memory T cells. Journal of immunology. 159:4611-9.
- 24. Aleksza, M, Lukacs A, Antal-Szalmas P, et al. 2002. Increased frequency of intracellular interleukin (IL)-13 and IL-10, but not IL-4, expressing CD4+ and CD8+ peripheral T cells of patients with atopic dermatitis. The British journal of dermatology. 147:1135-41.
- 25. La Grutta, S, Richiusa P, Pizzolanti G, et al. 2005. CD4(+)IL-13(+) cells in peripheral blood well correlates with the severity of atopic dermatitis in children. Allergy. 60:391-5.
- 26. Suárez-Fariñas, M, Dhingra N, Gittler J, et al. 2013. Intrinsic atopic dermatitis shows similar TH2 and higher TH17 immune activation compared with extrinsic atopic dermatitis. J Allergy Clin Immunol. 132:361-70.
- 27. Choy, DF, Hsu DK, Seshasayee D, et al. 2012. Comparative transcriptomic analyses of atopic dermatitis and psoriasis reveal shared neutrophilic inflammation. J Allergy Clin Immunol. 130:1335-43 e5.
- 28. Hamid, Q, Naseer T, Minshall EM, et al. 1996. In vivo expression of IL-12 and IL-13 in atopic dermatitis. J Allergy Clin Immunol. 98:225-31.
- 29. Jeong, CW, Ahn KS, Rho NK, et al. 2003. Differential in vivo cytokine mRNA expression in lesional skin of intrinsic vs. extrinsic atopic dermatitis patients using semiquantitative RT-PCR. Clin Exp Allergy. 33:1717-24.
- 30. Tazawa, T, Sugiura H, Sugiura Y, et al. 2004. Relative importance of IL-4 and IL-13 in lesional skin of atopic dermatitis. Archives of dermatological research. 295:459-64.
- 31. Neis, MM, Peters B, Dreuw A, et al. 2006. Enhanced expression levels of IL-31 correlate with IL-4 and IL-13 in atopic and allergic contact dermatitis. J Allergy Clin Immunol. 118:930-7.
- 32. Khattri, S, Shemer A, Rozenblit M, et al. 2014. Cyclosporine in patients with atopic dermatitis modulates activated inflammatory pathways and reverses epidermal pathology. J Allergy Clin Immunol. 133:1626-34.
- 33. Bunikowski, R, Staab D, Kussebi F, et al. 2001. Low-dose cyclosporin A microemulsion in children with severe atopic dermatitis: clinical and immunological effects. Pediatr Allergy Immunol. 12:216-23.
- 34. Tintle, S, Shemer A, Suarez-Farinas M, et al. 2011. Reversal of atopic dermatitis with narrow-band UVB phototherapy and biomarkers for therapeutic response. J Allergy Clin Immunol. 128:583-93 e1-4.
- 35. Wollenberg, A, Howell MD, Guttman-Yassky E, et al., editors. A Phase 2b Dose-Ranging Efficacy and Safety Study of Tralokinumab in Adult Patients with Moderate to Severe Atopic Dermatitis (AD). AAD 2017 2017; Orlando, FL.

DRM06-AD01-A2

36. Simpson, EL, Bieber T, Guttman-Yassky E, et al. 2016. Two Phase 3 Trials of Dupilumab versus Placebo in Atopic Dermatitis. The New England journal of medicine. 375:2335-48.

# 14 APPENDICES

Appendix 1. Schedule of Visits and Procedures

| Study Procedure | Screening | Baseline | Treatment Period | | | | | |
|---|---|---|---|---|---|---|---|---|
| Visit (V) | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 |
| Week (W) | -30 to -7 | W0 | W2 | W4 | W6 | W8 | W10 | W12 |
| Day (D)<br>Visit Window (d) | | D1 | D15 | D29 | D43 | D57 | D71 | D85 |
| Visit Willdow (d) | | | ±3d | ±3d | ±3d | ±3d | ±3d | ±3d |
| Screening/Baseline: | | | | | | | | |
| Informed Consent | Χ | | | | | | | |
| Inclusion/Exclusion | Χ | Х | | | | | | |
| Medical History/ Demographics | Χ | | | | | | | |
| Randomization | | Х | | | | | | |
| Safety: | | | | | | | | |
| Weight | Χ | Х | | | | | | |
| Height | Χ | | | | | | | |
| Vital Signs | Χ | Х | Χ | Χ | Χ | Х | Χ | Х |
| Physical Examination | X | | | | | | | |
| Adverse Events | | Х | Χ | X | X | Х | X | Х |
| Concomitant Medications | Χ | Х | Х | Х | Х | Х | Х | Х |
| Procedure/Therapy | Χ | Х | Х | Х | Х | Х | Χ | X |
| 12-Lead ECG | | Х | | | | | | |
| Laboratory Testing: | | | | | | | | |
| HIV Ab, HBsAg, HBcAb, Hep C<br>Ab | X | | | | | | | |
| Hematology, Chemistry | Х | Х | | Х | | Х | | Х |
| Urinalysis | Х | Х | | Х | | Х | | Х |
| Pregnancy Test (WOCBP only) | Serum | Urine | | Urine | | Urine | | Urine |
| Efficacy: | | | | | | | | |
| IGA | Χ | Х | | Х | | Х | | Х |
| EASI | Х | Х | | Х | | Х | | Х |
| BSA | Х | Х | | Х | | Х | | Х |
| Pruritus (daily) <sup>a</sup> | | Х | Х | Х | Х | Х | Х | Х |
| Sleep-loss (daily) a | | Х | Х | Х | Х | Х | Χ | Х |
| ADIQ <sup>a</sup> | | Х | Χ | Х | Х | Х | Χ | Х |
| POEM | | Х | | | | | | |
| DLQI | | Х | | | | Х | | |
| HADS | | Х | | | | Х | | |
| PK/Drug Concentration and Ar | nti-Drug Ant | ibody (ADA | A) Sample | es <sup>c</sup> : | | | | |
| PK Sample | | Х | Χ | X | | Х | | Х |
| ADA Sample | | Х | Х | Х | | | | |
| Treatment: | | | | | | | | |
| Administer Study Drug | | Х | Х | Χ | Х | Х | Х | Х |
| Reminders: | | | | | | | | |
| Apply emollient twice daily | | X | Х | Х | Χ | Х | Χ | X |
| Use electronic tablet daily | | X | Χ | Χ | Χ | X | Χ | X |

# Schedule of Visits and Procedures (cont'd)

| Study Procedure | | Treatment<br>Period | | Follow-up | /EOS | Unscheduled<br>Visit <sup>b</sup> | Early<br>Termination <sup>b</sup> |
|---|---|---|---|---|---|---|---|
| Visit (V) | V9 | V10 | V11 | V12 | V13 Phone<br>Call | | |
| Week (W) | W14 | W16 | W20 | W24 | W32 | | |
| Day (D) | D99 | D113 | D141 | D169 | D225 | | |
| Visit Window (d) | ±3d | ±3d | ±7d | ±7d | ±7d | | |
| Safety: | | ļ | | | | | |
| Weight | | Х | | | | | Х |
| Vital Signs | Х | Х | Х | Х | | Х | Х |
| Physical Examination | | Х | | | | | Х |
| Adverse Events | Х | Х | Х | Х | Х | Х | Х |
| Concomitant Medication | Х | Х | Х | Х | | Х | Х |
| Procedure/Therapy | Х | Х | Х | Х | | Х | Х |
| 12-Lead ECG | | Х | | | | | Х |
| Laboratory Testing: | | | | | | | |
| Hematology, Chemistry | 1 | Х | | Х | | | Х |
| Urinalysis | 1 | Х | | Х | | | Х |
| Pregnancy Test<br>(WOCBP only) | | Urine | | Urine | | | Urine |
| Efficacy: | | | | | | | |
| IGA | | Х | Х | Х | | | Х |
| EASI | | Х | X | X | | | X |
| BSA | | Х | X | Х | | | X |
| Pruritus (daily) a | Χ | X | | | | | X |
| Sleep-loss (daily) a | Χ | Х | | | | | X |
| ADIQ <sup>a</sup> | Х | Χ | | | | | X |
| POEM | | Х | | | | | Χ |
| DLQI | | Χ | | | | | Χ |
| HADS | | Х | | | | | X |
| Global Assessment of Change–AD | | X | | | | | X |
| PK/Drug Concentration | and Anti | -Drug Ar | ntibody (/ | ADA) Samp | oles <sup>c</sup> : | | |
| PK Sample | | Х | | Х | | | |
| ADA Sample | | Х | | Х | | | |
| Treatment: | | | | | | | |
| Administer Study Drug | Х | | | | | | |
| Reminders: | | | | | | | |
| Apply emollient twice daily | Х | Х | Х | Х | | | |
| Use electronic tablet daily a Pruritus NRS, sleep-lo | Х | | | | | | |

Pruritus NRS, sleep-loss NRS, and ADIQ are completed on an electronic tablet issued to the patient at the Baseline visit.

b If applicable.

<sup>&</sup>lt;sup>c</sup> PK and ADA samples taken pre-dose on dosing days (There is no dosing at the Week 16 and Week 24 visits).

# Appendix 2. Hanifin/Rajka Diagnostic Criteria for Atopic Dermatitis

From: Hanifin JM and Rajka G. Diagnostic features of atopic dermatitis. Acta Derm Venereol (Stockholm) 1980; Suppl 92:44–7.

To establish a diagnosis of atopic dermatitis the patient requires the presence of at least 3 "basic features" and 3 or more minor features listed below.

## **Basic Features**

Must have three or more basic features:

- Pruritus
- Typical morphology and distribution
- Flexural lichenification or linearity in adults
- Chronic or chronically-relapsing dermatitis
- Personal or family history of atopy (asthma, allergic rhinitis, atopic dermatitis)

### **Minor Features**

Plus, three or more minor features:

- Xerosis
- Ichthyosis, palmar hyperlinearity, or keratosis pilaris
- Immediate (type 1) skin-test reactivity
- Elevated serum IgE
- Early age of onset
- Tendency toward cutaneous infections (especially Staph. aureus and Herpes simplex)/impaired cell-mediated immunity
- Tendency toward non-specific hand or foot dermatitis
- Nipple eczema
- Cheilitis
- Recurrent conjunctivitis
- Dennie-Morgan infraorbital fold
- Keratoconus
- Anterior subcapsular cataracts
- Orbital darkening
- Facial pallor/facial erythema
- Pityriasis alba
- Anterior neck folds
- Itch when sweating
- Intolerance to wool and lipid solvents
- Perifollicular accentuation
- Food intolerance
- Course influenced by environmental or emotional factors
- White dermographism/delayed blanch

# Appendix 3. Investigator Global Assessment (IGA)

For IGA scoring, the Investigator should evaluate the patient's extent and severity of AD at a macroscopic level; i.e., without focusing on specific components of AD, which will be quantitated in the EASI score. In doing so, the investigator will use the table below to provide the IGA score.

| Score | Grade | Definition |
|---|---|---|
| 0 | Clear | Minor, residual discoloration; no erythema or induration/papulation; no oozing/crusting; no edema. |
| 1 | Almost Clear | Trace, faint pink erythema with barely perceptible induration/papulation and no oozing/crusting; no edema. |
| 2 | Mild | Faint-pink erythema with papulation and edema perceptible upon palpation and no oozing/crusting; minimal induration. |
| 3 | Moderate | Pink-red erythema with definite edema of skin papules and plaques; there may be some oozing/crusting; palpable induration. |
| 4 | Severe | Deep/bright red erythema with significant swelling and obvious raised borders of papules and plaques with oozing/crusting; significant induration. |





# Appendix 5. Body Surface Area (BSA)

The BSA assessment estimates the extent of disease or skin involvement with respect to AD and is expressed as a percentage of total body surface.

Determine BSA using the patient's palm = 1% rule.

The patient's palm is measured from the wrist to the proximal interphalangeal (PIP) and thumb.

Estimate the number of palms it takes to cover the affected AD area. Add up the number of palms to give a total estimate of the area covered in AD.

Below are estimates when entire areas (anterior and posterior) are covered:

Head and Neck = 10% (10 palms)

Upper Extremities = 20% (20 palms)

Trunk (axillae and groin) = 30% (30 palms)

Lower extremities (buttocks) = 40% (40 palms)

TOTAL BSA = 100% (100 palms)

#### Additional rules:

- 1. When many small lesions are present, try to put several together to make one patient palm.
- 2. Only include the edge of current lesions, not areas that have cleared.
- 3. Double check to see if area derived matches eyeball method.





| Appendix 8. | CCI |
|-------------|-----|

| 5. <mark>CC</mark> | | |
|--------------------|---------------------------------------|------|
| 6. | CI | |
| _ | • | |
| 7. | | |
| 8. | | |
| | | <br> |
| L | | |

| 9. | 9. CCI |
|----|----------------------|
| 10 | 10. CCI |
| | <del></del> |
| | 11. <mark>CCI</mark> |
| 11 | |
| 11 | |
| 11 | |
| 11 | |
| 11 | |
| 12 | |



# Appendix 9. Patient-Oriented Eczema Measure (POEM)

Please circle one response for each of the seven questions below about your eczema. Please leave blank any questions you feel unable to answer.

1. Over the last week, on how many days has your skin been itchy because of your eczema?

No davs

1-2 days

3-4 days

5–6 days

Every day

2. Over the last week, on how many nights has your sleep been disturbed because of your eczema?

No days

1-2 days

3-4 days

5–6 days

Every day

3. Over the last week, on how many days has your skin been bleeding because of your eczema?

No days

1–2 days

3-4 days

5-6 days

Every day

4. Over the last week, on how many days has your skin been weeping or oozing clear fluid because of your eczema?

No days

1–2 days

3–4 days

5–6 days

Every day

5. Over the last week, on how many days has your skin been cracked because of your eczema?

No days

1–2 days

3-4 days

5–6 days

Every day

6. Over the last week, on how many days has your skin been flaking off because of your eczema?

No days

1–2 days

3-4 days

5-6 days

Every day

7. Over the last week, on how many days has your skin felt dry or rough because of your eczema?

No days

1–2 days

3-4 days

5-6 days

Every day

Total POEM Score (Maximum 28): \_\_\_\_\_

# Appendix 10. Dermatology Life Quality Index (DLQI)

| The aim of this | questionnaire is to | measure how | much your s | kin problem l | has affected | your life |
|---|---|---|---|---|---|---|
| OVER THE LA | ST WEEK. Please | tick (X) one be | ox for each o | uestion. | | |

| 1. | Over the last week, how <b>itchy</b> , <b>sore</b> , <b>painful</b> or <b>stinging</b> has your skin been? | Very much<br>A lot<br>A little<br>Not at all | |
|---|---|---|---|
| 2. | Over the last week, how <b>embarrassed</b> or <b>self conscious</b> have you been because of your skin? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |
| 3. | Over the last week, how much has your skin interfered with you going <b>shopping</b> or looking after your <b>home</b> or <b>garden</b> ? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |
| 4. | Over the last week, how much has your skin influenced the <b>clothes</b> you wear? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |
| 5. | Over the last week, how much has your skin affected any <b>social</b> or <b>leisure</b> activities? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |
| 6. | Over the last week, how much has your skin made it difficult for you to do any <b>sport</b> ? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |
| 7. | Over the last week, has your skin prevented you from <b>working</b> or <b>studying</b> ? | Yes<br>No | |
| | If "No", over the last week how much has your skin been a problem at <b>work</b> or <b>studying</b> ? | A lot<br>A little<br>Not at all | |
| 8. | Over the last week, how much has your skin created problems with your <b>partner</b> or any of your <b>close friends</b> or <b>relatives</b> ? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |
| 9. | Over the last week, how much has your skin caused any sexual difficulties? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |
| 10. | Over the last week, how much of a problem has the <b>treatment</b> for your skin been, for example by making your home messy, or by taking up time? | Very much<br>A lot<br>A little<br>Not at all | Not relevant □ |

# DERMATOLOGY LIFE QUALITY INDEX (DLQI) - INSTRUCTIONS FOR USE

The Dermatology Life Quality Index questionnaire is designed for use in adults, i.e. patients over the age of 16. It is self-explanatory and can be simply handed to the patient who is asked to fill it in without the need for detailed explanation. It is usually completed in one or two minutes.

#### **SCORING**

The scoring of each question is as follows:

Very much Scored 3
A lot Scored 2
A little Scored 1
Not at all Scored 0
Not relevant Scored 0
Question 7, 'prevented work or studying' Scored 3

The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.

#### **HOW TO INTERPRET MEANING OF DLQI SCORES**

0–1 No effect at all on patient's life

2-5 Small effect on

patient's life

6–10 Moderate effect on

patient's life

11–20 Very large effect on

patient's life

21–30 Extremely large effect on patient's life

#### **REFERENCES**

Finlay AY and Khan GK. Dermatology Life Quality Index (DLQI): a simple practical measure for routine clinical use. *Clin Exp Dermatol* 1994; **19:**210-216.

Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. *Br J Dermatol* 2008; **159**:997-1035.

Hongbo Y, Thomas CL, Harrison MA, Salek MS, Finlay AY. Translating the science of quality of life into practice: What do dermatology life quality index scores mean? *J Invest Dermatol* 2005; **125**:659-64.

There is more information about the DLQI, including over 85 translations, at www.dermatology.org.uk. The DLQI is copyright but may be used without seeking permission by clinicians for routine clinical purposes. For other purposes, please contact the copyright owners.



# Appendix 12. Global Assessment of Change-AD

The following question will be asked at Week 16:

Overall, compared to the start of the study, how would you rate your atopic dermatitis symptoms over the past week?

- 1 = Much better
- 2 = Moderately better
- 3 = A little better
- 4 = No difference
- 5 = A little worse
- 6 = Moderately worse
- 7 = Much worse